CLINICAL TRIAL: NCT02294734
Title: A Randomised, Double-blind (Sponsor Unblinded), Placebo-controlled, Parallel-group, Multicentre Study to Evaluate the Efficacy and Safety of GSK2269557 Administered in Addition to Standard of Care in Adult Subjects Diagnosed With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: An Efficacy Study of GSK2269557 Added to Standard Care in Subjects With an Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116678; 2014-001972-70 (EudraCT Number)
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: functional respiratory capacity; High-resolution computed tomography; GSK2269557; acute exacerbation of COPD; lung capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nemiralisib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2269557 repeat dose (Experimental): Participants will receive 2 inhalation of GSK2269557 dry powder once daily via DISKUS™ 'device' (DISKUS is a trademark of the GSK group of companies)
  Interventions: Drug: GSK2269557
- Matching placebo repeat dose (Placebo Comparator): Participants will receive 2 inhalation matching placebo dry powder once daily via DISKUS 'device'
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2269557 — Dry powder for inhalation via DISKUS 'device' with unit dose strength of 500 micrograms (mcg) per actuation with total dose of 1000 mcg daily
  Arms: GSK2269557 repeat dose
Drug: Placebo — Dry powder for inhalation via DISKUS 'device'
  Arms: Matching placebo repeat dose

SUMMARY:
The purpose of this study is to evaluate the efficacy of GSK2269557 administered in addition to standard of care in adult subjects diagnosed with an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD). Additionally study will also assess safety, tolerability and pharmacokinetic data. The total duration of the study will be 13-14 weeks including screening, treatment period and a follow up visit. Subjects will receive once daily study treatment administration starting on Day 1. Study is planned to recruit approximately 120 subjects such that approximately 100 subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years of age inclusive, at the time of signing the informed consent
* The subject has a confirmed and established diagnosis of COPD, as defined by the global initiative for chronic Obstructive Lung Disease (GOLD) guidelines for at least 6 months prior to entry.
* The subject has a post-bronchodilator FEV1/Forced Vital Capacity (FVC) < 0.7 and FEV1 <= 80 % of predicted (Predictions should be according to the European Community of Coal and Steel [ECCS] equations), documented in the last 5 years.
* Disease severity: Acute exacerbation of COPD requiring an escalation in therapy to include corticosteroid and antibiotics. Acute exacerbation to be confirmed by an experienced physician and represent a recent change in at least two major and one minor symptoms, one major and two minor symptoms, or all 3 major symptoms. Major symptoms: subjective increase in dyspnea, increase in sputum volume, and change in sputum colour. Minor symptoms: cough, wheeze and sore throat.
* The subject is a smoker or an ex-smoker with a smoking history of at least 10 pack years (pack years = [cigarettes per day smoked/20 x number of years smoked])
* Body weight >= 45 kilogram (kg) and body mass index (BMI) within the range 18 - 32 kg/metered squared (m^2) (inclusive).
* Male
* Female subject : is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as: Pre-menopausal females with one of the following: documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy and documented bilateral oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until completion of the follow-up visit.

GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP):

Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label.

Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label.

Oral Contraceptive, either combined or progestogen alone. Injectable progestogen. Contraceptive vaginal ring. Percutaneous contraceptive patches. Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.

Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository).

* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until after the completion of the follow up visit.

Vasectomy with documentation of azoospermia. Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label. Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label. Oral Contraceptive, either combined or progestogen alone or injectable progestogen. Contraceptive vaginal ring. Percutaneous contraceptive patches.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the study protocol.

Exclusion Criteria:

* To avoid recruitment of subjects with a severe COPD exacerbation, the presence of any one of the following severity criteria will render the subject ineligible for inclusion in the study:

Need for invasive mechanical ventilation (short term (< 48hour) Non-invasive Ventilation (NIV) or Continuous Positive Airway Pressure [CPAP] is acceptable).

Haemodynamic instability or clinically significant heart failure. Confusion.

* Subjects who have a history or current medical conditions or diseases that are not well controlled and, which as judged by the Investigator, may affect subject safety or influence the outcome of the study. (Note: Patients with adequately treated and well controlled concurrent medical conditions [e.g. hypertension or non-insulin dependent diabetes mellitus] are permitted to be entered into the study).
* Subject has a diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, pulmonary fibrosis, asthma or any other respiratory condition that might, in the opinion of the investigator, compromise the safety of the subject or affect the interpretation of the results.
* Alanine aminotransferase >2x upper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the exclusion criteria, outside of the reference range for the population being studied may be included if the Investigator [in consultation with the GSK Medical Monitor if required] documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* ECG indicative of an acute cardiac event (e.g. Myocardial Infarction) or demonstrating a clinically significant arrhythmia requiring treatment.
* QTcF > 450 millisecond (msec) or QTcF > 480 msec in subjects with Bundle Branch Block, based on single QTcF value.
* Subjects who have undergone lung volume reduction surgery.
* Subject is currently on chronic treatment with macrolides; long term oxygen therapy (> 15 hours/day).
* The subject has been on chronic treatment with anti-Tumour Necrosis Factor (anti-TNF), anti-Interleukin-1 (anti-IL1), or any other immunosuppressive therapy within 60 days prior to dosing.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >28 units for males or >21 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint ( equivalent to 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof (such as lactose) or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* A known (historical) positive test for human immune virus (HIV) antibody.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. NOTE: Because of the short window for screening, treatment with GSK2269557 may start before receiving the result of the hepatitis tests. If subsequently the test is found to be positive, the subject may be withdrawn, as judged by the Principal Investigator in consultation with the Medical Monitor.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-02-19 (Actual); Study Completion 2016-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Belgium (2):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Erpent
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense
- Netherlands (3):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Zutphen
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Timișoara
- Russia (6):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Vladimir
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20859

REFERENCES:
- [Background] Cahn A, Hamblin JN, Robertson J, Begg M, Jarvis E, Wilson R, Dear G, Leemereise C, Cui Y, Mizuma M, Montembault M, Van Holsbeke C, Vos W, De Backer W, De Backer J, Hessel EM. An Inhaled PI3Kdelta Inhibitor Improves Recovery in Acutely Exacerbating COPD Patients: A Randomized Trial. Int J Chron Obstruct Pulmon Dis. 2021 Jun 3;16:1607-1619. doi: 10.2147/COPD.S309129. eCollection 2021. PMID 34113093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a screening visit, a 12-week treatment period, and a 1-2 week post-treatment follow-up. The total duration of the study was 13-14 weeks including the screening visit.
Pre-assignment Details: Approximately 120 participants with an acute exacerbation of chronic obstructive pulmonary disease (COPD) were randomized (1:1) to GSK 2269557 1000 micrograms (µg) and placebo such that approximately 100 participants complete the study. Participants were also stratified by whether they were willing and able to provide sputum samples at screening.
Groups:
- Placebo: Participants received placebo two inhalations per day administered via a dry powder inhaler for a duration of 84 days.
- GSK2269557 1000 mcg: Participants received 1000 mcg of GSK2269557 two inhalations per day administered via a dry powder inhaler for a duration of 84 days.
Period: Overall Study
Arm/Group | Placebo | GSK2269557 1000 mcg
Started | 63 | 63
Completed | 49 | 55
Not Completed | 14 | 8
Not completed — Adverse Event | 5 | 5
Not completed — Met Protocol Defined Stopping Criteria | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2269557 1000 mcg | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (7.88) | 65.6 (7.14) | 65.2 (7.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 46 | 46 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Specific Imaging Airway Volume (siVaw), Measured at FRC and TLC Scan Conditions, Presented in Longitudinal and Scan Trimmed Scan Types, Measured in 5 Lobes and 5 Regions at Screening, Day 12 and Day 28
Description: siVaw is a measure of the volume in an individual's airway corrected for their lobar volume derived from the high resolution computed tomography (HRCT). It was measured at functional residual volume (FRC) and total lung capacity (TLC). Data was collected at longitudinal time points: Screening, Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (RUL, LUL, RML, RLL & LLL) and 5 Regions (Upper, Lower, Central, Distal & Total). For longitudinal time points and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only particpants available at the specified time point were analysed (represented by n=X1, X2 in the category title).
Time Frame: Baseline, Day 12 and Day 28
Population: Intention to Treat (ITT) Population excluding the subject with a pacemaker.
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliter/Liter (mL/L)
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 62 | 63
Milliliter/Liter (mL/L)
  FRC; Longitudinal; Lobes; RUL; D12 , n =54, 57 | 1.033 [0.851 to 1.255] | 1.052 [0.924 to 1.197]
  FRC; Longitudinal; Lobes; RUL; D28 , n =56, 56 | 0.983 [0.775 to 1.246] | 1.075 [0.940 to 1.230]
  FRC; Longitudinal; Lobes; LUL; D12 , n=56, 59 | 0.975 [0.817 to 1.165] | 1.000 [0.877 to 1.140]
  FRC; Longitudinal; Lobes; LUL; D28 , n =56, 58 | 0.893 [0.745 to 1.070] | 1.090 [0.932 to 1.275]
  FRC; Longitudinal; Lobes; RML; D12 , n =52, 58 | 0.956 [0.806 to 1.135] | 0.871 [0.691 to 1.097]
  FRC; Longitudinal; Lobes; RML; D28 , n=53, 57 | 0.853 [0.677 to 1.075] | 1.006 [0.867 to 1.167]
  FRC; Longitudinal; Lobes; RLL; D12 , n =54, 59 | 0.908 [0.684 to 1.204] | 1.115 [0.885 to 1.405]
  FRC; Longitudinal; Lobes; RLL; D28 , n =55, 58 | 0.871 [0.652 to 1.164] | 1.167 [0.975 to 1.397]
  FRC; Longitudinal; Lobes; LLL; D12 , n =53, 58 | 1.051 [0.885 to 1.248] | 1.087 [0.892 to 1.323]
  FRC; Longitudinal; Lobes; LLL; D28 ,n =54, 58 | 1.000 [0.806 to 1.242] | 1.199 [0.999 to 1.438]
  FRC; Scan Trimmed; Lobes; RUL; SCRD12 , n =54, 57 | 1.049 [0.956 to 1.151] | 1.002 [0.921 to 1.090]
  FRC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 56 | 0.999 [0.892 to 1.118] | 0.993 [0.910 to 1.083]
  FRC; Scan Trimmed; Lobes; RUL; D12D28 , n =51, 55 | 0.931 [0.858 to 1.010] | 0.995 [0.933 to 1.062]
  FRC; Scan Trimmed; Lobes; LUL; SCRD12 , n =56, 59 | 0.979 [0.891 to 1.077] | 1.012 [0.938 to 1.092]
  FRC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 58 | 0.952 [0.862 to 1.051] | 1.018 [0.934 to 1.110]
  FRC; Scan Trimmed; Lobes; LUL; D12D28 , n =53, 57 | 0.973 [0.893 to 1.061] | 1.014 [0.942 to 1.090]
  FRC; Scan Trimmed; Lobes; RML; SCRD12 , n =52, 58 | 0.924 [0.811 to 1.052] | 0.977 [0.878 to 1.087]
  FRC; Scan Trimmed; Lobes; RML; SCRD28 , n=53, 57 | 0.927 [0.832 to 1.034] | 0.967 [0.872 to 1.073]
  FRC; Scan Trimmed; Lobes; RML; D12D28 , n =52, 56 | 0.927 [0.830 to 1.035] | 1.023 [0.925 to 1.131]
  FRC; Scan Trimmed; Lobes; RLL; SCRD12 , n =54, 59 | 0.987 [0.863 to 1.129] | 1.000 [0.893 to 1.121]
  FRC; Scan Trimmed; Lobes; RLL; SCRD28 , n=55, 58 | 0.972 [0.815 to 1.159] | 1.014 [0.916 to 1.121]
  FRC; Scan Trimmed; Lobes; RLL; D12D28 , n =52, 57 | 0.920 [0.829 to 1.020] | 1.015 [0.918 to 1.121]
  FRC; Scan Trimmed; Lobes; LLL; SCRD12 , n =53, 58 | 1.031 [0.925 to 1.149] | 1.050 [0.939 to 1.173]
  FRC; Scan Trimmed; Lobes; LLL; SCRD28 , n=54, 58 | 1.034 [0.893 to 1.198] | 1.064 [0.958 to 1.180]
  FRC; Scan Trimmed; Lobes; LLL; D12D28 , n =51, 56 | 0.978 [0.897 to 1.066] | 1.055 [0.953 to 1.168]
  FRC; Longitudinal;Region; Upper; D12 , n =56, 59 | 0.952 [0.809 to 1.120] | 1.004 [0.891 to 1.132]
  FRC; Longitudinal; Region; Upper; D28 , n =56, 58 | 0.918 [0.769 to 1.096] | 1.066 [0.939 to 1.210]
  FRC; Longitudinal; Region; Lower; D12 , n=54, 59 | 0.989 [0.819 to 1.194] | 1.065 [0.878 to 1.291]
  FRC; Longitudinal; Region; Lower; D28 , n =55, 58 | 0.952 [0.772 to 1.172] | 1.150 [0.979 to 1.351]
  FRC; Longitudinal; Region;Central; D12 , n =56, 59 | 0.969 [0.886 to 1.060] | 1.021 [0.963 to 1.083]
  FRC; Longitudinal;Region; Central; D28 , n=56, 58 | 0.992 [0.918 to 1.071] | 1.002 [0.958 to 1.050]
  FRC; Longitudinal; Region; Distal; D12 , n =56, 59 | 0.963 [0.801 to 1.158] | 1.027 [0.889 to 1.188]
  FRC; Longitudinal; Region; Distal D28 , n =56, 58 | 0.939 [0.778 to 1.134] | 1.098 [0.959 to 1.258]
  FRC; Longitudinal; Region;Total; D12, n =56, 59 | 0.970 [0.881 to 1.068] | 1.018 [0.955 to 1.085]
  FRC; Longitudinal; Region; Total; D28 ,n =56, 58 | 0.989 [0.911 to 1.074] | 1.009 [0.959 to 1.061]
  FRC; Scan Trimmed; Region;Upper; SCRD12 ,n =56, 59 | 0.989 [0.899 to 1.088] | 1.001 [0.929 to 1.078]
  FRC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 58 | 0.962 [0.878 to 1.054] | 1.007 [0.925 to 1.096]
  FRC; Scan Trimmed; Region;Upper; D12D28 ,n =53, 57 | 0.967 [0.889 to 1.051] | 1.011 [0.949 to 1.077]
  FRC; Scan Trimmed; Region;Lower; SCRD12 ,n =54, 59 | 1.019 [0.920 to 1.128] | 1.028 [0.924 to 1.145]
  FRC; Scan Trimmed; Region; Lower; SCRD28 ,n=55, 58 | 1.002 [0.868 to 1.157] | 1.039 [0.944 to 1.144]
  FRC; Scan Trimmed; Region;Lower; D12D28 ,n =52, 57 | 0.953 [0.873 to 1.040] | 1.008 [0.920 to 1.104]
  FRC;Scan Trimmed;Region;Central; SCRD12 ,n =56, 59 | 0.988 [0.911 to 1.072] | 1.022 [0.964 to 1.084]
  FRC;Scan Trimmed; Region Central; SCRD28 ,n=56, 58 | 1.002 [0.932 to 1.078] | 0.999 [0.954 to 1.047]
  FRC;Scan Trimmed;Region Central; D12D28 ,n =53, 57 | 0.998 [0.942 to 1.057] | 0.977 [0.932 to 1.025]
  FRC;Scan Trimmed; Region;Distal; SCRD12 ,n =56, 59 | 0.998 [0.903 to 1.104] | 1.009 [0.925 to 1.099]
  FRC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 58 | 0.984 [0.883 to 1.095] | 1.021 [0.936 to 1.115]
  FRC;Scan Trimmed;Region;Distal; D12D28 , n =53, 57 | 0.963 [0.887 to 1.044] | 1.019 [0.950 to 1.092]
  FRC;Scan Trimmed; Region;Total; SCRD12 , n =56, 59 | 0.989 [0.911 to 1.074] | 1.019 [0.960 to 1.082]
  FRC;Scan Trimmed;Region;Total; SCRD28 , n=56, 58 | 1.002 [0.931 to 1.078] | 1.000 [0.953 to 1.049]
  Trimmed;Region;Total; D12D28 , n =53, 57 | 0.995 [0.940 to 1.054] | 0.982 [0.936 to 1.030]
  TLC; Longitudinal; Lobes; RUL; D12 , n =58, 57 | 1.048 [0.951 to 1.154] | 0.976 [0.912 to 1.043]
  TLC; Longitudinal; Lobes; RUL; D28 , n =56, 57 | 1.045 [0.927 to 1.179] | 0.979 [0.908 to 1.055]
  TLC; Longitudinal; Lobes; LUL; D12 , n=58, 59 | 1.043 [0.933 to 1.166] | 1.007 [0.936 to 1.083]
  TLC; Longitudinal; Lobes; LUL; D28 , n =56, 59 | 1.078 [0.922 to 1.260] | 1.027 [0.947 to 1.115]
  TLC; Longitudinal; Lobes; RML; D12 , n =57, 58 | 1.087 [0.906 to 1.304] | 0.894 [0.787 to 1.016]
  TLC; Longitudinal; Lobes; RML; D28 , n=56, 58 | 1.084 [0.893 to 1.317] | 0.903 [0.808 to 1.008]
  TLC; Longitudinal; Lobes; RLL; D12 , n =58, 59 | 1.038 [0.884 to 1.219] | 0.906 [0.820 to 1.001]
  TLC; Longitudinal; Lobes; RLL; D28 , n =56, 59 | 1.014 [0.839 to 1.227] | 0.948 [0.858 to 1.048]
  TLC; Longitudinal; Lobes; LLL; D12 , n =57, 59 | 1.074 [0.917 to 1.258] | 0.934 [0.844 to 1.035]
  TLC; Longitudinal; Lobes; LLL; D28 ,n =55, 59 | 1.075 [0.901 to 1.282] | 0.993 [0.891 to 1.107]
  TLC; Scan Trimmed; Lobes; RUL; SCRD12 , n =58, 57 | 1.040 [0.978 to 1.105] | 0.988 [0.940 to 1.038]
  TLC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 57 | 1.020 [0.949 to 1.097] | 0.981 [0.925 to 1.040]
  TLC; Scan Trimmed; Lobes; RUL; D12D28 , n =55, 56 | 0.971 [0.908 to 1.039] | 1.002 [0.956 to 1.050]
  TLC; Scan Trimmed; Lobes; LUL; SCRD12 , n =58, 59 | 1.022 [0.961 to 1.088] | 1.001 [0.950 to 1.055]
  TLC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 59 | 1.035 [0.962 to 1.113] | 0.991 [0.933 to 1.052]
  TLC; Scan Trimmed; Lobes; LUL; D12D28 , n =55, 58 | 1.007 [0.933 to 1.086] | 1.002 [0.956 to 1.050]
  TLC; Scan Trimmed; Lobes; RML; SCRD12 , n =57, 58 | 1.029 [0.948 to 1.116] | 0.934 [0.870 to 1.003]
  TLC; Scan Trimmed; Lobes; RML; SCRD28 , n=56, 58 | 1.020 [0.933 to 1.116] | 0.932 [0.877 to 0.991]
  TLC; Scan Trimmed; Lobes; RML; D12D28 , n =55, 57 | 0.980 [0.904 to 1.063] | 1.008 [0.942 to 1.078]
  TLC; Scan Trimmed; Lobes; RLL; SCRD12 , n =58, 59 | 1.022 [0.940 to 1.112] | 0.932 [0.871 to 0.996]
  TLC; Scan Trimmed; Lobes; RLL; SCRD28 , n=56, 59 | 0.984 [0.897 to 1.078] | 0.944 [0.884 to 1.008]
  TLC; Scan Trimmed; Lobes; RLL; D12D28 , n =55, 58 | 0.962 [0.881 to 1.051] | 1.027 [0.980 to 1.076]
  TLC; Scan Trimmed; Lobes; LLL; SCRD12 , n =57, 59 | 1.024 [0.939 to 1.117] | 0.967 [0.908 to 1.030]
  TLC; Scan Trimmed; Lobes; LLL; SCRD28 , n=55, 59 | 1.025 [0.933 to 1.125] | 0.972 [0.907 to 1.043]
  TLC; Scan Trimmed; Lobes; LLL; D12D28 , n =54, 58 | 0.984 [0.911 to 1.062] | 1.017 [0.970 to 1.065]
  TLC; Longitudinal;Region; Upper; D12 , n =58, 59 | 1.031 [0.935 to 1.137] | 0.983 [0.922 to 1.049]
  TLC; Longitudinal; Region; Upper; D28 , n =56, 59 | 1.046 [0.918 to 1.191] | 0.995 [0.928 to 1.067]
  TLC; Longitudinal; Region; Lower; D12 , n=58, 59 | 1.051 [0.909 to 1.215] | 0.924 [0.840 to 1.017]
  TLC; Longitudinal; Region; Lower; D28 , n =56, 59 | 1.037 [0.879 to 1.223] | 0.974 [0.883 to 1.074]
  TLC; Longitudinal; Region;Central; D12 , n =58, 59 | 1.001 [0.971 to 1.033] | 0.991 [0.971 to 1.012]
  TLC; Longitudinal;Region; Central; D28 , n=56, 59 | 1.006 [0.979 to 1.033] | 0.992 [0.972 to 1.013]
  TLC; Longitudinal; Region; Distal; D12 , n =58, 59 | 1.043 [0.931 to 1.168] | 0.949 [0.883 to 1.021]
  TLC; Longitudinal; Region; Distal D28 , n =56, 59 | 1.039 [0.902 to 1.197] | 0.982 [0.910 to 1.060]
  TLC; Longitudinal; Region;Total; D12, n =58, 59 | 1.009 [0.969 to 1.051] | 0.982 [0.958 to 1.006]
  TLC; Longitudinal; Region; Total; D28 ,n =56, 59 | 1.005 [0.967 to 1.044] | 0.988 [0.964 to 1.013]
  TLC; Scan Trimmed; Region;Upper; SCRD12 ,n =58, 59 | 1.028 [0.969 to 1.090] | 0.992 [0.944 to 1.041]
  TLC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 59 | 1.021 [0.953 to 1.095] | 0.984 [0.932 to 1.040]
  TLC; Scan Trimmed; Region;Upper; D12D28 ,n =55, 58 | 0.985 [0.922 to 1.054] | 1.003 [0.962 to 1.046]
  TLC; Scan Trimmed; Region;Lower; SCRD12 ,n =58, 59 | 1.021 [0.943 to 1.105] | 0.954 [0.897 to 1.014]
  TLC; Scan Trimmed; Region; Lower; SCRD28 ,n=56, 59 | 0.996 [0.916 to 1.083] | 0.960 [0.899 to 1.025]
  TLC; Scan Trimmed; Region;Lower; D12D28 ,n =55, 58 | 0.972 [0.899 to 1.052] | 1.018 [0.977 to 1.060]
  TLC;Scan Trimmed;Region;Central; SCRD12 ,n =58, 59 | 1.000 [0.972 to 1.029] | 0.997 [0.975 to 1.020]
  TLC;Scan Trimmed; Region Central; SCRD28 ,n=56, 59 | 1.005 [0.981 to 1.030] | 0.995 [0.972 to 1.018]
  TLC;Scan Trimmed;Region Central; D12D28 ,n =55, 58 | 1.004 [0.981 to 1.028] | 0.998 [0.984 to 1.012]
  TLC;Scan Trimmed; Region;Distal; SCRD12 ,n =58, 59 | 1.025 [0.960 to 1.095] | 0.972 [0.922 to 1.025]
  TLC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 59 | 1.008 [0.936 to 1.086] | 0.972 [0.919 to 1.029]
  TLC;Scan Trimmed;Region;Distal; D12D28 , n =55, 58 | 0.978 [0.912 to 1.050] | 1.011 [0.973 to 1.051]
  TLC;Scan Trimmed; Region;Total; SCRD12 , n =58, 59 | 1.005 [0.973 to 1.037] | 0.991 [0.967 to 1.017]
  TLC;Scan Trimmed;Region;Total; SCRD28 , n=56, 59 | 1.004 [0.976 to 1.032] | 0.989 [0.965 to 1.014]
  TLC; Scan Trimmed;Region;Total; D12D28 , n =55, 58 | 0.997 [0.970 to 1.025] | 1.000 [0.984 to 1.017]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 60.66, Bayesian repeated measures model — The data entered for the p-value represents the posterior probability that the true treatment ratio is greater than 1. P-value is denoted in percentage; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted, accounting for correlation within region and visit; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.85 to 1.25] — FRC; Longitudinal; Lobes; RUL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.21, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.19, 95% CI 2-sided [0.97 to 1.47] — FRC; Longitudinal; Lobes; RUL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 74.29, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.88 to 1.28] — FRC; Longitudinal; Lobes; LUL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.48, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.29, 95% CI 2-sided [1.06 to 1.58] — FRC; Longitudinal; Lobes; LUL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 5: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 13.98, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.87, 95% CI 2-sided [0.66 to 1.13] — FRC; Longitudinal; Lobes; RML; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 6: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.92, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.28, 95% CI 2-sided [1.01 to 1.62] — FRC; Longitudinal; Lobes; RML; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 7: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 80.24, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.14, 95% CI 2-sided [0.84 to 1.54] — FRC; Longitudinal; Lobes; RLL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 8: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.79, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.30, 95% CI 2-sided [1.01 to 1.66] — FRC; Longitudinal; Lobes; RLL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 9: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 51.27, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.81 to 1.25] — FRC; Longitudinal; Lobes; LLL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 10: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 90.66, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.15, 95% CI 2-sided [0.93 to 1.42] — FRC; Longitudinal; Lobes; LLL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 11: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 54.89, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.90 to 1.12] — FRC; Scan Trimmed; Lobes; RUL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 12: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.45, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.10, 95% CI 2-sided [0.98 to 1.24] — FRC; Scan Trimmed; Lobes; RUL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 13: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.09, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.09, 95% CI 2-sided [0.98 to 1.21] — FRC; Scan Trimmed; Lobes; RUL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 14: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 62.95, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.91 to 1.14] — FRC; Scan Trimmed; Lobes; LUL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 15: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.86, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.12, 95% CI 2-sided [0.99 to 1.26] — FRC; Scan Trimmed; Lobes; LUL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 16: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.16, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.09, 95% CI 2-sided [0.98 to 1.20] — FRC; Scan Trimmed; Lobes; LUL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 17: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 48.99, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.86 to 1.15] — FRC; Scan Trimmed; Lobes; RML; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 18: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.51, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.12, 95% CI 2-sided [0.98 to 1.28] — FRC; Scan Trimmed; Lobes; RML; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 19: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.59, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.13, 95% CI 2-sided [0.97 to 1.31] — FRC; Scan Trimmed; Lobes; RML; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 20: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 61.27, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.86 to 1.23] — FRC; Scan Trimmed; Lobes; RLL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 21: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.63, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; Non-informative priors used for all modelling parameters. Unstructured covariance matrix fitted, accounting for correlation within region and visit.No; Posterior Median Ratio = 1.15, 95% CI 2-sided [0.99 to 1.34] — FRC; Scan Trimmed; Lobes; RLL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 22: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.02, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.12, 95% CI 2-sided [0.97 to 1.29] — FRC; Scan Trimmed; Lobes; RLL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 23: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 53.24, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.87 to 1.17] — FRC; Scan Trimmed; Lobes; LLL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 24: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 70.84, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.91 to 1.19] — FRC; Scan Trimmed; Lobes; LLL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 25: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 74.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.92 to 1.19] — FRC; Scan Trimmed; Lobes; LLL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 26: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 65.43, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.87 to 1.24] — FRC; Longitudinal;Region; Upper; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 27: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.19, 95% CI 2-sided [0.99 to 1.42] — FRC; Longitudinal; Region; Upper; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 28: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.99, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.81 to 1.34] — FRC; Longitudinal; Region; Lower; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 29: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 91.99, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.15, 95% CI 2-sided [0.94 to 1.41] — FRC; Longitudinal; Region; Lower; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 30: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 76.81, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.94 to 1.14] — FRC; Longitudinal; Region;Central; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 31: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 67.01, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.95 to 1.09] — FRC; Longitudinal;Region; Central; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 32: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.91, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.85 to 1.27] — FRC; Longitudinal; Region; Distal; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 33: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.47, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.18, 95% CI 2-sided [0.99 to 1.42] — FRC; Longitudinal; Region; Distal D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 34: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 72.17, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.93 to 1.14] — FRC; Longitudinal; Region;Total; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 35: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 74.38, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.95 to 1.11] — FRC; Longitudinal; Region; Total; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 36: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 53.85, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.90 to 1.12] — FRC; Scan Trimmed; Region;Upper; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 37: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.02, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.10, 95% CI 2-sided [0.98 to 1.23] — FRC; Scan Trimmed; Region;Upper; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 38: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 92.27, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.97 to 1.18] — FRC; Scan Trimmed; Region;Upper; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 39: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 54.65, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.88 to 1.16] — FRC; Scan Trimmed; Region;Lower; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 40: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 87.93, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.95 to 1.23] — FRC; Scan Trimmed; Region; Lower; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 41: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 77.57, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.92 to 1.19] — FRC; Scan Trimmed; Region;Lower; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 42: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 77.07, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.95 to 1.11] — FRC;Scan Trimmed;Region;Central; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 43: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 78.42, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.96 to 1.10] — FRC;Scan Trimmed; Region Central; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 44: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 44.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.93 to 1.06] — FRC;Scan Trimmed;Region Central; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 45: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 52.79, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.89 to 1.13] — FRC;Scan Trimmed; Region;Distal; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 46: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.51, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.10, 95% CI 2-sided [0.98 to 1.24] — FRC;Scan Trimmed;Region; Distal; SCRD28 .The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 47: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 93.16, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.98 to 1.19] — FRC;Scan Trimmed;Region;Distal; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 48: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 73.70, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.95 to 1.11] — FRC;Scan Trimmed; Region;Total; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 49: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 81.04, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.96 to 1.10] — FRC;Scan Trimmed;Region;Total; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 50: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 52.58, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.94 to 1.07] — FRC; Scan Trimmed;Region;Total; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 51: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 15.85, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.86 to 1.05] — TLC; Longitudinal; Lobes; RUL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 52: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 48.69, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.90 to 1.11] — TLC; Longitudinal; Lobes; RUL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 53: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 52.25, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.90 to 1.13] — TLC; Longitudinal; Lobes; LUL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 54: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 66.48, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.91 to 1.16] — TLC; Longitudinal; Lobes; LUL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 55: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.12, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.88, 95% CI 2-sided [0.72 to 1.06] — TLC; Longitudinal; Lobes; RML; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 56: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 16.95, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.78 to 1.09] — TLC; Longitudinal; Lobes; RML; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 57: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.89, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.75 to 1.05] — TLC; Longitudinal; Lobes; RLL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 58: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 50.40, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.86 to 1.17] — TLC; Longitudinal; Lobes; RLL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 59: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 7.44, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.76 to 1.04] — TLC; Longitudinal; Lobes; LLL; D12 .The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 60: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 56.35, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.87 to 1.18] — TLC; Longitudinal; Lobes; LLL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 61: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 4.03, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.93, 95% CI 2-sided [0.87 to 1.01] — TLC; Scan Trimmed; Lobes; RUL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 62: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 24.79, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.89 to 1.06] — TLC; Scan Trimmed; Lobes; RUL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 63: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 77.08, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.95 to 1.12] — TLC; Scan Trimmed; Lobes; RUL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 64: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 23.07, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.89 to 1.05] — TLC; Scan Trimmed; Lobes; LUL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 65: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 18.58, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.88 to 1.05] — TLC; Scan Trimmed; Lobes; LUL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 66: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 44.94, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.92 to 1.08] — TLC; Scan Trimmed; Lobes; LUL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 67: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 2.21, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.80 to 1.00] — TLC; Scan Trimmed; Lobes; RML; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 68: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 6.09, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.83 to 1.02] — TLC; Scan Trimmed; Lobes; RML; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 69: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 66.60, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.92 to 1.13] — TLC; Scan Trimmed; Lobes; RML; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 70: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 3.23, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.90, 95% CI 2-sided [0.81 to 1.01] — TLC; Scan Trimmed; Lobes; RLL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 71: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 20.83, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.86 to 1.07] — TLC; Scan Trimmed; Lobes; RLL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 72: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 87.60, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.96 to 1.16] — TLC; Scan Trimmed; Lobes; RLL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 73: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 7.90, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.93, 95% CI 2-sided [0.84 to 1.03] — TLC; Scan Trimmed; Lobes; LLL; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 74: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 23.39, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.87 to 1.07] — TLC; Scan Trimmed; Lobes; LLL; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 75: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 76.16, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.95 to 1.12] — TLC; Scan Trimmed; Lobes; LLL; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 76: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 22.54, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.87 to 1.06] — TLC; Longitudinal;Region; Upper; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 77: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 58.17, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.91 to 1.12] — TLC; Longitudinal; Region; Upper; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 78: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 6.22, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.76 to 1.03] — TLC; Longitudinal; Region; Lower; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 79: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 55.85, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.88 to 1.17] — TLC; Longitudinal; Region; Lower; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 80: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 25.44, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.02] — TLC; Longitudinal; Region;Central; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 81: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 18.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.02] — TLC; Longitudinal;Region; Cetral; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 82: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 8.12, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.82 to 1.04] — TLC; Longitudinal; Region; Distal; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 83: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 57.39, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.90 to 1.13] — TLC; Longitudinal; Region; Distal D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 84: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 10.00, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.93 to 1.02] — TLC; Longitudinal; Region;Total; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 85: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 29.88, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.95 to 1.03] — TLC; Longitudinal; Region; Total; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 86: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 12.63, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.89 to 1.03] — TLC; Scan Trimmed; Region;Upper; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 87: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 32.29, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.91 to 1.06] — TLC; Scan Trimmed; Region;Upper; SCRD28 The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 88: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 69.92, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.95 to 1.10] — TLC; Scan Trimmed; Region;Upper; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 89: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 6.10, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.93, 95% CI 2-sided [0.84 to 1.02] — TLC; Scan Trimmed; Region;Lower; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 90: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 33.63, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.89 to 1.08] — TLC; Scan Trimmed; Region; Lower; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 91: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 86.07, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.97 to 1.13] — TLC; Scan Trimmed; Region;Lower; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 92: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 41.38, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.96 to 1.03] — TLC;Scan Trimmed;Region;Central; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 93: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 24.88, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.02] — TLC;Scan Trimmed; Region Central; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 94: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 29.89, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.97 to 1.02] — TLC;Scan Trimmed;Region Central; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 95: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 7.13, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.94, 95% CI 2-sided [0.87 to 1.02] — TLC;Scan Trimmed; Region;Distal; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 96: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 32.91, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.90 to 1.07] — TLC;Scan Trimmed;Region; Distal; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 97: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 81.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.96 to 1.11] — TLC;Scan Trimmed;Region;Distal; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 98: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 21.87, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.95 to 1.02] — TLC;Scan Trimmed; Region;Total; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 99: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 24.49, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.95 to 1.02] — TLC;Scan Trimmed;Region;Total; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 100: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 55.52, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.97 to 1.03] — TLC; Scan Trimmed;Region;Total; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval

2. Secondary Outcome: Change From Baseline in Imaging Airways Volume: iVaw, Measured at FRC and TLC Scan Conditions, Presented in Longitudinal and Scan Trimmed Scan Types, Measured in 5 Lobes and 5 Regions at Screening, Day 12 and Day 28
Description: iVaw was derived from HRCT to evaluate the effect of once daily inhaled dose of GSK2269557 on lung parameters. Data was collected at longitudinal time points: Screening, Day 12 & Day 28 and at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (RUL, LUL, RML, RLL & LLL) and 5 Regions (Upper, Lower, Central, Distal & Total). For longitudinal time points and SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only particpants available at the specified time point were analysed (represented by n=X1, X2 in the category title).
Time Frame: Baseline, Day 12 and Day 28
Population: ITT Population excluding the subject with a pacemaker.
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliter (mL)
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 62 | 63
Milliliter (mL)
  FRC; Longitudinal; Lobes; RUL; D12 , n =54, 59 | 1.020 [0.838 to 1.242] | 1.058 [0.930 to 1.203]
  FRC; Longitudinal; Lobes; RUL; D28 , n =56, 58 | 0.960 [0.755 to 1.220] | 1.121 [0.965 to 1.301]
  FRC; Longitudinal; Lobes; LUL; D12 , n=56, 59 | 0.951 [0.789 to 1.145] | 0.999 [0.866 to 1.151]
  FRC; Longitudinal; Lobes; LUL; D28 , n =56, 58 | 0.876 [0.727 to 1.055] | 1.108 [0.938 to 1.309]
  FRC; Longitudinal; Lobes; RML; D12 , n =53, 59 | 0.905 [0.746 to 1.098] | 0.869 [0.694 to 1.089]
  FRC; Longitudinal; Lobes; RML; D28 , n=53, 58 | 0.835 [0.655 to 1.064] | 1.013 [0.870 to 1.180]
  FRC; Longitudinal; Lobes; RLL; D12 , n =54, 59 | 0.889 [0.669 to 1.182] | 1.119 [0.892 to 1.404]
  FRC; Longitudinal; Lobes; RLL; D28 , n =55, 58 | 0.850 [0.634 to 1.140] | 1.177 [0.977 to 1.417]
  FRC; Longitudinal; Lobes; LLL; D12 , n =53, 58 | 1.017 [0.853 to 1.212] | 1.067 [0.881 to 1.293]
  FRC; Longitudinal; Lobes; LLL; D28 ,n =54, 58 | 0.980 [0.784 to 1.226] | 1.187 [0.992 to 1.421]
  FRC; Scan Trimmed; Lobes; RUL; SCRD12 , n =54, 59 | 1.035 [0.942 to 1.137] | 1.006 [0.927 to 1.091]
  FRC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 58 | 0.976 [0.872 to 1.091] | 1.027 [0.938 to 1.124]
  FRC; Scan Trimmed; Lobes; RUL; D12D28 , n =51, 57 | 0.927 [0.861 to 0.997] | 1.018 [0.948 to 1.092]
  FRC; Scan Trimmed; Lobes; LUL; SCRD12 , n =56, 59 | 0.954 [0.870 to 1.048] | 1.010 [0.932 to 1.095]
  FRC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 58 | 0.933 [0.846 to 1.029] | 1.035 [0.946 to 1.133]
  FRC; Scan Trimmed; Lobes; LUL; D12D28 , n =53, 57 | 0.981 [0.902 to 1.068] | 1.029 [0.956 to 1.107]
  FRC; Scan Trimmed; Lobes; RML; SCRD12 , n =53, 59 | 0.905 [0.798 to 1.027] | 0.970 [0.872 to 1.079]
  FRC; Scan Trimmed; Lobes; RML; SCRD28 , n=53, 58 | 0.907 [0.807 to 1.020] | 0.972 [0.876 to 1.079]
  FRC; Scan Trimmed; Lobes; RML; D12D28 , n =52, 57 | 0.927 [0.833 to 1.032] | 1.031 [0.933 to 1.139]
  FRC; Scan Trimmed; Lobes; RLL; SCRD12 , n =54, 59 | 0.968 [0.849 to 1.102] | 1.004 [0.905 to 1.113]
  FRC; Scan Trimmed; Lobes; RLL; SCRD28 , n=55, 58 | 0.948 [0.796 to 1.131] | 1.022 [0.925 to 1.130]
  FRC; Scan Trimmed; Lobes; RLL; D12D28 , n =52, 57 | 0.916 [0.837 to 1.002] | 1.018 [0.920 to 1.125]
  FRC; Scan Trimmed; Lobes; LLL; SCRD12 , n =53, 58 | 0.997 [0.898 to 1.108] | 1.031 [0.935 to 1.136]
  FRC; Scan Trimmed; Lobes; LLL; SCRD28 , n=54, 58 | 1.013 [0.869 to 1.182] | 1.054 [0.954 to 1.164]
  FRC; Scan Trimmed; Lobes; LLL; D12D28 , n =51, 56 | 0.989 [0.922 to 1.061] | 1.061 [0.962 to 1.170]
  FRC; Longitudinal;Region; Upper; D12 , n =56, 59 | 0.933 [0.789 to 1.104] | 1.000 [0.882 to 1.133]
  FRC; Longitudinal; Region; Upper; D28 , n =56, 58 | 0.898 [0.749 to 1.077] | 1.079 [0.943 to 1.236]
  FRC; Longitudinal; Region; Lower; D12 , n=54, 59 | 0.965 [0.798 to 1.166] | 1.058 [0.878 to 1.275]
  FRC; Longitudinal; Region; Lower; D28 , n =55, 58 | 0.931 [0.751 to 1.153] | 1.151 [0.978 to 1.354]
  FRC; Longitudinal; Region;Central; D12 , n =56, 59 | 0.945 [0.863 to 1.035] | 1.016 [0.961 to 1.074]
  FRC; Longitudinal;Region; Cetral; D28 , n=56, 58 | 0.968 [0.892 to 1.050] | 1.010 [0.961 to 1.062]
  FRC; Longitudinal; Region; Distal; D12 , n =56, 59 | 0.939 [0.779 to 1.132] | 1.022 [0.883 to 1.182]
  FRC; Longitudinal; Region; Distal D28 , n =56, 58 | 0.917 [0.757 to 1.110] | 1.107 [0.961 to 1.276]
  FRC; Longitudinal; Region;Total; D12 n =56, 59 | 0.946 [0.858 to 1.043] | 1.012 [0.951 to 1.077]
  FRC; Longitudinal; Region; Total; D28 ,n =56, 58 | 0.966 [0.885 to 1.053] | 1.017 [0.961 to 1.076]
  FRC; Scan Trimmed; Region;Upper; SCRD12 ,n =56, 59 | 0.969 [0.881 to 1.067] | 0.997 [0.923 to 1.076]
  FRC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 58 | 0.941 [0.860 to 1.030] | 1.019 [0.934 to 1.112]
  FRC; Scan Trimmed; Region;Upper; D12D28 ,n =53, 57 | 0.968 [0.893 to 1.049] | 1.025 [0.960 to 1.095]
  FRC; Scan Trimmed; Region;Lower; SCRD12 ,n =54, 59 | 0.994 [0.902 to 1.096] | 1.022 [0.929 to 1.124]
  FRC; Scan Trimmed; Region; Lower; SCRD28 ,n=55, 58 | 0.980 [0.846 to 1.135] | 1.040 [0.948 to 1.140]
  FRC; Scan Trimmed; Region;Lower; D12D28 ,n =52, 57 | 0.954 [0.889 to 1.02] | 1.013 [0.928 to 1.106]
  FRC;Scan Trimmed;Region;Central; SCRD12 ,n =56, 59 | 0.964 [0.891 to 1.044] | 1.016 [0.967 to 1.069]
  FRC;Scan Trimmed; Region Central; SCRD28 ,n=56, 58 | 0.978 [0.908 to 1.054] | 1.007 [0.966 to 1.051]
  FRC;Scan Trimmed;Region Central; D12D28 ,n =53, 57 | 1.000 [0.950 to 1.053] | 0.988 [0.946 to 1.033]
  FRC;Scan Trimmed; Region;Distal; SCRD12 ,n =56, 59 | 0.974 [0.882 to 1.074] | 1.003 [0.923 to 1.089]
  FRC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 58 | 0.960 [0.862 to 1.070] | 1.030 [0.944 to 1.123]
  FRC;Scan Trimmed;Region;Distal; D12D28 , n =53, 57 | 0.965 [0.897 to 1.039] | 1.030 [0.961 to 1.105]
  FRC;Scan Trimmed; Region;Total; SCRD12 , n =56, 59 | 0.965 [0.891 to 1.045] | 1.014 [0.963 to 1.067]
  FRC;Scan Trimmed;Region;Total; SCRD28 , n=56, 58 | 0.978 [0.908 to 1.054] | 1.008 [0.964 to 1.053]
  FRC; Scan Trimmed;Region;Total; D12D28 , n =53, 57 | 0.998 [0.949 to 1.049] | 0.993 [0.949 to 1.039]
  TLC; Longitudinal; Lobes; RUL; D12 , n =58, 59 | 1.057 [0.954 to 1.172] | 0.982 [0.917 to 1.051]
  TLC; Longitudinal; Lobes; RUL; D28 , n =56, 59 | 1.050 [0.920 to 1.198] | 0.989 [0.916 to 1.068]
  TLC; Longitudinal; Lobes; LUL; D12 , n=58, 59 | 1.045 [0.929 to 1.175] | 1.005 [0.932 to 1.084]
  TLC; Longitudinal; Lobes; LUL; D28 , n =56, 59 | 1.082 [0.913 to 1.282] | 1.025 [0.942 to 1.116]
  TLC; Longitudinal; Lobes; RML; D12 , n =58, 59 | 1.045 [0.861 to 1.268] | 0.887 [0.779 to 1.009]
  TLC; Longitudinal; Lobes; RML; D28 , n=56, 59 | 1.076 [0.872 to 1.328] | 0.906 [0.810 to 1.012]
  TLC; Longitudinal; Lobes; RLL; D12 , n =58, 59 | 1.049 [0.889 to 1.238] | 0.910 [0.817 to 1.014]
  TLC; Longitudinal; Lobes; RLL; D28 , n =56, 59 | 1.014 [0.826 to 1.244] | 0.956 [0.854 to 1.071]
  TLC; Longitudinal; Lobes; LLL; D12, n =57, 59 | 1.082 [0.911 to 1.286] | 0.924 [0.827 to 1.031]
  TLC; Longitudinal; Lobes; LLL; D28 ,n =55, 59 | 1.077 [0.888 to 1.306] | 0.989 [0.879 to 1.112]
  TLC; Scan Trimmed; Lobes; RUL; SCRD12 , n =58, 59 | 1.049 [0.982 to 1.121] | 0.994 [0.945 to 1.046]
  TLC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 59 | 1.025 [0.944 to 1.113] | 0.987 [0.932 to 1.046]
  TLC; Scan Trimmed; Lobes; RUL; D12D28 , n =55, 58 | 0.966 [0.898 to 1.039] | 1.002 [0.957 to 1.050]
  TLC; Scan Trimmed; Lobes; LUL; SCRD12 , n =58, 59 | 1.024 [0.958 to 1.095] | 0.999 [0.946 to 1.055]
  TLC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 59 | 1.039 [0.954 to 1.132] | 0.989 [0.929 to 1.052]
  TLC; Scan Trimmed; Lobes; LUL; D12D28 , n =55, 58 | 1.008 [0.929 to 1.095] | 1.002 [0.957 to 1.049]
  TLC; Scan Trimmed; Lobes; RML; SCRD12 , n =58, 59 | 1.017 [0.937 to 1.105] | 0.926 [0.861 to 0.996]
  TLC; Scan Trimmed; Lobes; RML; SCRD28 , n=56, 59 | 1.013 [0.915 to 1.121] | 0.935 [0.879 to 0.995]
  TLC; Scan Trimmed; Lobes; RML; D12D28 , n =55, 58 | 0.974 [0.898 to 1.057] | 1.021 [0.955 to 1.090]
  TLC; Scan Trimmed; Lobes; RLL; SCRD12 , n =58, 59 | 1.032 [0.947 to 1.126] | 0.936 [0.875 to 1.001]
  TLC; Scan Trimmed; Lobes; RLL; SCRD28 , n=56, 59 | 0.983 [0.884 to 1.094] | 0.952 [0.892 to 1.016]
  TLC; Scan Trimmed; Lobes; RLL; D12D28 , n =55, 58 | 0.953 [0.868 to 1.047] | 1.033 [0.986 to 1.082]
  TLC; Scan Trimmed; Lobes; LLL; SCRD12 , n =57, 59 | 1.032 [0.940 to 1.133] | 0.956 [0.895 to 1.022]
  TLC; Scan Trimmed; Lobes; LLL; SCRD28 , n=55, 59 | 1.027 [0.919 to 1.147] | 0.968 [0.904 to 1.037]
  TLC; Scan Trimmed; Lobes; LLL; D12D28 , n =54, 58 | 0.976 [0.906 to 1.052] | 1.025 [0.976 to 1.077]
  TLC; Longitudinal;Region; Upper; D12 , n =58, 59 | 1.037 [0.934 to 1.151] | 0.981 [0.917 to 1.049]
  TLC; Longitudinal; Region; Upper; D28 , n =56, 59 | 1.049 [0.909 to 1.211] | 0.994 [0.924 to 1.069]
  TLC; Longitudinal; Region; Lower; D12 , n=58, 59 | 1.061 [0.911 to 1.235] | 0.921 [0.830 to 1.022]
  TLC; Longitudinal; Region; Lower; D28 , n =56, 59 | 1.037 [0.867 to 1.241] | 0.977 [0.876 to 1.089]
  TLC; Longitudinal; Region;Central; D12 , n =58, 59 | 1.006 [0.972 to 1.042] | 0.988 [0.970 to 1.007]
  TLC; Longitudinal;Region; Cetral; D28 , n=56, 59 | 1.007 [0.968 to 1.049] | 0.993 [0.973 to 1.013]
  TLC; Longitudinal; Region; Distal; D12 , n =58, 59 | 1.048 [0.930 to 1.182] | 0.947 [0.876 to 1.023]
  TLC; Longitudinal; Region; Distal D28 , n =56, 59 | 1.041 [0.891 to 1.215] | 0.983 [0.905 to 1.067]
  TLC; Longitudinal; Region;Total; D12, n =58, 59 | 1.014 [0.968 to 1.062] | 0.979 [0.954 to 1.004]
  TLC; Longitudinal; Region; Total; D28 ,n =56, 59 | 1.007 [0.955 to 1.061] | 0.989 [0.963 to 1.016]
  TLC; Scan Trimmed; Region;Upper; SCRD12 ,n =58, 59 | 1.033 [0.969 to 1.102] | 0.989 [0.940 to 1.041]
  TLC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 59 | 1.025 [0.945 to 1.111] | 0.983 [0.929 to 1.040]
  TLC; Scan Trimmed; Region;Upper; D12D28 ,n =55, 58 | 0.983 [0.915 to 1.055] | 1.006 [0.964 to 1.049]
  TLC; Scan Trimmed; Region;Lower; SCRD12 ,n =58, 59 | 1.030 [0.949 to 1.118] | 0.951 [0.894 to 1.011]
  TLC; Scan Trimmed; Region; Lower; SCRD28 ,n=56, 59 | 0.997 [0.904 to 1.099] | 0.963 [0.903 to 1.027]
  TLC; Scan Trimmed; Region;Lower; D12D28 ,n =55, 58 | 0.964 [0.889 to 1.045] | 1.025 [0.985 to 1.067]
  TLC;Scan Trimmed;Region;Central; SCRD12 ,n =58, 59 | 1.005 [0.973 to 1.037] | 0.994 [0.976 to 1.013]
  TLC;Scan Trimmed; Region Central; SCRD28 ,n=56, 59 | 1.007 [0.971 to 1.044] | 0.995 [0.977 to 1.014]
  TLC;Scan Trimmed;Region Central; D12D28 ,n =55, 58 | 1.000 [0.980 to 1.022] | 1.003 [0.991 to 1.015]
  TLC;Scan Trimmed; Region;Distal; SCRD12 ,n =58, 59 | 1.030 [0.961 to 1.105] | 0.969 [0.918 to 1.023]
  TLC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 59 | 1.010 [0.927 to 1.100] | 0.973 [0.919 to 1.030]
  TLC;Scan Trimmed;Region;Distal; D12D28 , n =55, 58 | 0.975 [0.906 to 1.04] | 1.016 [0.978 to 1.057]
  TLC;Scan Trimmed; Region;Total; SCRD12 , n =58, 59 | 1.010 [0.974 to 1.046] | 0.989 [0.967 to 1.011]
  TLC;Scan Trimmed;Region;Total; SCRD28 , n=56, 59 | 1.006 [0.966 to 1.047] | 0.990 [0.968 to 1.012]
  TLC; Scan Trimmed;Region;Total; D12D28 , n =55, 58 | 0.993 [0.968 to 1.019] | 1.005 [0.990 to 1.020]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 59.55, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.84 to 1.25] — (FRC; Longitudinal; Lobes; RUL; D12, The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.01, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.18, 95% CI 2-sided [0.96 to 1.46] — (FRC; Longitudinal; Lobes; RUL; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 82.27, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.10, 95% CI 2-sided [0.90 to 1.33] — FRC; Longitudinal; Lobes; LUL; D12, The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.22, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.31, 95% CI 2-sided [1.06 to 1.61] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 46.24, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.75 to 1.29] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.30, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.29, 95% CI 2-sided [1.02 to 1.64] — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 92.60, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.25, 95% CI 2-sided [0.92 to 1.70] — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.01, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.38, 95% CI 2-sided [1.05 to 1.81] — [estimate comment as in outcome 1, analysis 8]
Statistical Analysis 9: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 58.80, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.82 to 1.28] — [estimate comment as in outcome 1, analysis 9]
Statistical Analysis 10: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 86.82, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.13, 95% CI 2-sided [0.91 to 1.42] — [estimate comment as in outcome 1, analysis 10]
Statistical Analysis 11: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 67.37, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.92 to 1.14] — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 12: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.35, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.14, 95% CI 2-sided [1.01 to 1.29] — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 13: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.86, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.10, 95% CI 2-sided [0.99 to 1.23] — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 14: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 86.18, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.95 to 1.19] — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 15: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.89, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.16, 95% CI 2-sided [1.02 to 1.31] — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 16: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 91.94, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.97 to 1.19] — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 17: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 55.32, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.88 to 1.17] — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 18: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.17, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.15, 95% CI 2-sided [1.00 to 1.32] — [estimate comment as in outcome 1, analysis 18]
Statistical Analysis 19: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.57, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.14, 95% CI 2-sided [0.99 to 1.32] — [estimate comment as in outcome 1, analysis 19]
Statistical Analysis 20: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 79.13, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.90 to 1.27] — [estimate comment as in outcome 1, analysis 20]
Statistical Analysis 21: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.54, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.22, 95% CI 2-sided [1.05 to 1.42] — [estimate comment as in outcome 1, analysis 21]
Statistical Analysis 22: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.80, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.14, 95% CI 2-sided [1.00 to 1.30] — [estimate comment as in outcome 1, analysis 22]
Statistical Analysis 23: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 71.94, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.91 to 1.19] — [estimate comment as in outcome 1, analysis 23]
Statistical Analysis 24: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 85.30, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.94 to 1.23] — [estimate comment as in outcome 1, analysis 24]
Statistical Analysis 25: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 82.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.94 to 1.19] — [estimate comment as in outcome 1, analysis 25]
Statistical Analysis 26: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 72.55, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.88 to 1.27] — [estimate comment as in outcome 1, analysis 26]
Statistical Analysis 27: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.44, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.22, 95% CI 2-sided [1.02 to 1.47] — [estimate comment as in outcome 1, analysis 27]
Statistical Analysis 28: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 78.24, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.11, 95% CI 2-sided [0.86 to 1.43] — [estimate comment as in outcome 1, analysis 28]
Statistical Analysis 29: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.80, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.23, 95% CI 2-sided [0.99 to 1.52] — [estimate comment as in outcome 1, analysis 29]
Statistical Analysis 30: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 91.11, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.97 to 1.17] — [estimate comment as in outcome 1, analysis 30]
Statistical Analysis 31: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 89.30, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.97 to 1.13] — FRC; Longitudinal;Region; Cetral; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 32: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 74.67, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.87 to 1.32] — [estimate comment as in outcome 1, analysis 32]
Statistical Analysis 33: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.25, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.23, 95% CI 2-sided [1.02 to 1.48] — [estimate comment as in outcome 1, analysis 33]
Statistical Analysis 34: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 87.80, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.96 to 1.18] — [estimate comment as in outcome 1, analysis 34]
Statistical Analysis 35: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 91.54, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.97 to 1.15] — [estimate comment as in outcome 1, analysis 35]
Statistical Analysis 36: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 68.89, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.92 to 1.14] — [estimate comment as in outcome 1, analysis 36]
Statistical Analysis 37: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.19, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.13, 95% CI 2-sided [1.01 to 1.27] — [estimate comment as in outcome 1, analysis 37]
Statistical Analysis 38: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.07, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.98 to 1.19] — [estimate comment as in outcome 1, analysis 38]
Statistical Analysis 39: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.74, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.92 to 1.19] — [estimate comment as in outcome 1, analysis 39]
Statistical Analysis 40: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.83, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.12, 95% CI 2-sided [0.99 to 1.28] — [estimate comment as in outcome 1, analysis 40]
Statistical Analysis 41: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 79.80, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.94 to 1.17] — [estimate comment as in outcome 1, analysis 41]
Statistical Analysis 42: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.29, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.99 to 1.13] — FRC;Scan Trimmed;Region;Central; SCRD12 .The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 43: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.27, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.99 to 1.13] — [estimate comment as in outcome 1, analysis 43]
Statistical Analysis 44: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 47.62, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.94 to 1.06] — [estimate comment as in outcome 1, analysis 44]
Statistical Analysis 45: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 71.55, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.92 to 1.15] — [estimate comment as in outcome 1, analysis 45]
Statistical Analysis 46: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.29, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.13, 95% CI 2-sided [1.01 to 1.28] — FRC;Scan Trimmed;Region; Distal; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 47: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.09, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Bayesian repeated measures model = 1.08, 95% CI 2-sided [0.99 to 1.19] — [estimate comment as in outcome 1, analysis 47]
Statistical Analysis 48: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 93.68, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.98 to 1.13] — [estimate comment as in outcome 1, analysis 48]
Statistical Analysis 49: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.58, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [1.00 to 1.14] — [estimate comment as in outcome 1, analysis 49]
Statistical Analysis 50: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 56.99, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.95 to 1.06] — [estimate comment as in outcome 1, analysis 50]
Statistical Analysis 51: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 13.08, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.94, 95% CI 2-sided [0.85 to 1.04] — [estimate comment as in outcome 1, analysis 51]
Statistical Analysis 52: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 52.99, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.89 to 1.13] — [estimate comment as in outcome 1, analysis 52]
Statistical Analysis 53: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 60.75, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.90 to 1.14] — [estimate comment as in outcome 1, analysis 53]
Statistical Analysis 54: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.23, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.92 to 1.20] — [estimate comment as in outcome 1, analysis 54]
Statistical Analysis 55: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 28.14, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.78 to 1.14] — [estimate comment as in outcome 1, analysis 55]
Statistical Analysis 56: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 38.43, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.84 to 1.14] — [estimate comment as in outcome 1, analysis 56]
Statistical Analysis 57: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 25.21, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.80 to 1.12] — [estimate comment as in outcome 1, analysis 57]
Statistical Analysis 58: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 81.73, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.91 to 1.27] — [estimate comment as in outcome 1, analysis 58]
Statistical Analysis 59: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.87, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.90, 95% CI 2-sided [0.76 to 1.06] — TLC; Longitudinal; Lobes; LLL; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 60: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.87 to 1.21] — [estimate comment as in outcome 1, analysis 60]
Statistical Analysis 61: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 4.03, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.93, 95% CI 2-sided [0.86 to 1.01] — [estimate comment as in outcome 1, analysis 61]
Statistical Analysis 62: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 30.03, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.89 to 1.07] — [estimate comment as in outcome 1, analysis 62]
Statistical Analysis 63: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 80.34, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.95 to 1.13] — [estimate comment as in outcome 1, analysis 63]
Statistical Analysis 64: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 25.65, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.89 to 1.06] — [estimate comment as in outcome 1, analysis 64]
Statistical Analysis 65: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 24.36, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.88 to 1.06] — [estimate comment as in outcome 1, analysis 65]
Statistical Analysis 66: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 48.45, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.91 to 1.09] — [estimate comment as in outcome 1, analysis 66]
Statistical Analysis 67: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 1.95, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.81 to 0.99] — [estimate comment as in outcome 1, analysis 67]
Statistical Analysis 68: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 14.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.94, 95% CI 2-sided [0.85 to 1.05] — [estimate comment as in outcome 1, analysis 68]
Statistical Analysis 69: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 80.61, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.95 to 1.16] — [estimate comment as in outcome 1, analysis 69]
Statistical Analysis 70: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 3.30, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.91, 95% CI 2-sided [0.81 to 1.01] — TLC; Scan Trimmed; Lobes; RLL; SCRD12.The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 71: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 42.22, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.88 to 1.11] — [estimate comment as in outcome 1, analysis 71]
Statistical Analysis 72: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.24, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.09, 95% CI 2-sided [0.99 to 1.20] — TLC; Scan Trimmed; Lobes; RLL; D12D28The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 73: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 6.38, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.83 to 1.03] — [estimate comment as in outcome 1, analysis 73]
Statistical Analysis 74: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 28.82, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.86 to 1.09] — [estimate comment as in outcome 1, analysis 74]
Statistical Analysis 75: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 87.39, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.05, 95% CI 2-sided [0.97 to 1.14] — [estimate comment as in outcome 1, analysis 75]
Statistical Analysis 76: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 23.27, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.87 to 1.07] — TLC; Longitudinal; Region; Upper; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 77: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 57.82, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.90 to 1.13] — TLC; Longitudinal; Region; Upper; D28.The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 78: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.67, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.90, 95% CI 2-sided [0.77 to 1.06] — [estimate comment as in outcome 1, analysis 78]
Statistical Analysis 79: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 70.73, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.89 to 1.22] — [estimate comment as in outcome 1, analysis 79]
Statistical Analysis 80: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 25.61, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.95 to 1.02] — TLC; Longitudinal; Region; Central; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 81: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 44.10, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.96 to 1.03] — TLC; Longitudinal; Region; Cetral; D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 82: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 10.14, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.82 to 1.04] — [estimate comment as in outcome 1, analysis 82]
Statistical Analysis 83: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 62.87, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.90 to 1.16] — [estimate comment as in outcome 1, analysis 83]
Statistical Analysis 84: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 11.82, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.93 to 1.02] — TLC; Longitudinal; Region; Total; D12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 85: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 51.44, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.95 to 1.05] — [estimate comment as in outcome 1, analysis 85]
Statistical Analysis 86: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.54, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.88 to 1.03] — TLC; Scan Trimmed; Region; Upper; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 87: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 30.03, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.89 to 1.07] — TLC; Scan Trimmed; Region; Upper; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 88: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 73.03, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.95 to 1.11] — TLC; Scan Trimmed; Region; Upper; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 89: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 4.64, Bayesian repeated measures model. — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.83 to 1.01] — TLC; Scan Trimmed; Region; Lower; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 90: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 42.13, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.89 to 1.10] — [estimate comment as in outcome 1, analysis 90]
Statistical Analysis 91: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 93.33, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.98 to 1.16] — TLC; Scan Trimmed; Region; Lower; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 92: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 27.33, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.95 to 1.02] — TLC; Scan Trimmed; Region; Central; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 93: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 34.15, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.03] — TLC; Scan Trimmed; Region Central; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 94: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 58.42, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.98 to 1.03] — TLC; Scan Trimmed; Region Central; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 95: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 5.93, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.94, 95% CI 2-sided [0.86 to 1.02] — TLC; Scan Trimmed; Region; Distal; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 96: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 35.88, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.89 to 1.08] — TLC; Scan Trimmed; Region; Distal; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 97: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 86.41, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.97 to 1.13] — TLC; Scan Trimmed; Region; Distal; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 98: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 13.52, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.94 to 1.02] — TLC; Scan Trimmed; Region; Total; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 99: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 32.84, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.95 to 1.03] — TLC; Scan Trimmed; Region; Total; SCRD28 .The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 100: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 78.09, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.98 to 1.04] — TLC; Scan Trimmed; Region; Total; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval

3. Secondary Outcome: Change From Baseline in Imaging Airways Resistance ( iRaw) Measured at FRC and TLC Scan Conditions, Presented in Scan Trimmed Scan Types, Measured in 5 Lobes and 5 Regions at Screening, Day 12 and Day 28
Description: iRaw was derived from HRCT to evaluate the effect of once daily inhaled dose of GSK2269557 on lung parameters. It was measured at functional residual volume (FRC) and total lung capacity (TLC). Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (RUL, LUL, RML, RLL & LLL) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only particpants available at the specified time point were analysed (represented by n=X1, X2 in the category title).
Time Frame: Baseline, Day 12 and Day 28
Population: ITT Population excluding the subject with a pacemaker.
Measure: Geometric Mean (95% Confidence Interval); unit: Kilopascal (Kpa)*s/L
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 62 | 63
Kilopascal (Kpa)*s/L
  FRC; Scan Trimmed; Lobes; RUL; SCRD12 , n =54, 59 | 0.908 [0.620 to 1.330] | 0.948 [0.693 to 1.296]
  FRC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 58 | 0.849 [0.529 to 1.362] | 0.958 [0.701 to 1.309]
  FRC; Scan Trimmed; Lobes; RUL; D12D28 , n =51, 57 | 1.039 [0.715 to 1.510] | 0.898 [0.697 to 1.157]
  FRC; Scan Trimmed; Lobes; LUL; SCRD12 , n =56, 59 | 0.982 [0.687 to 1.403] | 0.946 [0.706 to 1.267]
  FRC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 58 | 0.937 [0.620 to 1.417] | 0.820 [0.568 to 1.186]
  FRC; Scan Trimmed; Lobes; LUL; D12D28 , n =53, 57 | 0.842 [0.603 to 1.176] | 0.934 [0.703 to 1.241]
  FRC; Scan Trimmed; Lobes; RML; SCRD12 , n =53, 59 | 1.022 [0.667 to 1.568] | 0.998 [0.656 to 1.520]
  FRC; Scan Trimmed; Lobes; RML; SCRD28 , n=53, 58 | 1.378 [0.865 to 2.196] | 0.886 [0.632 to 1.240]
  FRC; Scan Trimmed; Lobes; RML; D12D28 , n =52, 57 | 1.027 [0.692 to 1.523] | 1.198 [0.811 to 1.769]
  FRC; Scan Trimmed; Lobes; RLL; SCRD12 , n =54, 59 | 1.100 [0.705 to 1.716] | 1.043 [0.673 to 1.617]
  FRC; Scan Trimmed; Lobes; RLL; SCRD28 , n=55, 58 | 1.504 [1.011 to 2.237] | 1.044 [0.728 to 1.497]
  FRC; Scan Trimmed; Lobes; RLL; D12D28 , n =52, 57 | 1.289 [0.953 to 1.745] | 1.126 [0.773 to 1.641]
  FRC; Scan Trimmed; Lobes; LLL; SCRD12 , n =53, 58 | 0.781 [0.522 to 1.167] | 0.738 [0.491 to 1.109]
  FRC; Scan Trimmed; Lobes; LLL; SCRD28 , n=54, 58 | 0.949 [0.637 to 1.414] | 0.818 [0.546 to 1.227]
  FRC; Scan Trimmed; Lobes; LLL; D12D28 , n =51, 56 | 1.051 [0.818 to 1.350] | 1.012 [0.700 to 1.465]
  FRC; Scan Trimmed; Region;Upper; SCRD12 ,n =56, 59 | 0.934 [0.656 to 1.329] | 0.960 [0.735 to 1.255]
  FRC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 58 | 0.940 [0.629 to 1.404] | 0.887 [0.643 to 1.222]
  FRC; Scan Trimmed; Region;Upper; D12D28 ,n =53, 57 | 0.869 [0.617 to 1.223] | 1.127 [0.834 to 1.52]
  FRC; Scan Trimmed; Region;Lower; SCRD12 ,n =54, 59 | 0.845 [0.543 to 1.314] | 0.821 [0.531 to 1.270]
  FRC; Scan Trimmed; Region; Lower; SCRD28 ,n=55, 58 | 1.215 [0.835 to 1.766] | 0.868 [0.606 to 1.243]
  FRC; Scan Trimmed; Region;Lower; D12D28 ,n =52, 57 | 1.113 [0.887 to 1.396] | 1.193 [0.805 to 1.766]
  FRC;Scan Trimmed;Region;Central; SCRD12 ,n =56, 59 | 1.104 [0.832 to 1.464] | 0.933 [0.769 to 1.133]
  FRC;Scan Trimmed; Region Central; SCRD28 ,n=56, 58 | 1.079 [0.794 to 1.465] | 0.950 [0.810 to 1.114]
  FRC;Scan Trimmed;Region Central; D12D28 ,n =53, 57 | 1.033 [0.851 to 1.253] | 1.010 [0.854 to 1.195]
  FRC;Scan Trimmed; Region;Distal; SCRD12 ,n =56, 59 | 0.800 [0.546 to 1.174] | 0.859 [0.600 to 1.230]
  FRC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 58 | 0.993 [0.675 to 1.459] | 0.873 [0.636 to 1.199]
  FRC;Scan Trimmed;Region;Distal; D12D28 , n =53, 57 | 0.887 [0.670 to 1.175] | 1.220 [0.890 to 1.674]
  FRC;Scan Trimmed; Region;Total; SCRD12 , n =56, 59 | 1.006 [0.760 to 1.333] | 0.919 [0.738 to 1.145]
  FRC;Scan Trimmed;Region;Total; SCRD28 , n=56, 58 | 1.036 [0.758 to 1.417] | 0.922 [0.750 to 1.132]
  FRC; Scan Trimmed;Region;Total; D12D28 , n =53, 57 | 1.000 [0.820 to 1.220] | 1.066 [0.875 to 1.298]
  TLC; Scan Trimmed; Lobes; RUL; SCRD12 , n =56, 59 | 0.843 [0.677 to 1.049] | 0.978 [0.810 to 1.181]
  TLC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 58 | 0.929 [0.714 to 1.210] | 1.019 [0.826 to 1.258]
  TLC; Scan Trimmed; Lobes; RUL; D12D28 , n =53, 57 | 1.152 [0.953 to 1.391] | 0.901 [0.759 to 1.069]
  TLC; Scan Trimmed; Lobes; LUL; SCRD12 , n =56, 59 | 0.879 [0.717 to 1.077] | 0.979 [0.829 to 1.156]
  TLC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 58 | 0.922 [0.726 to 1.173] | 0.886 [0.687 to 1.141]
  TLC; Scan Trimmed; Lobes; LUL; D12D28 , n =53, 57 | 1.025 [0.857 to 1.226] | 0.894 [0.750 to 1.066]
  TLC; Scan Trimmed; Lobes; RML; SCRD12 , n =57, 58 | 1.076 [0.834 to 1.388] | 1.349 [1.001 to 1.816]
  TLC; Scan Trimmed; Lobes; RML; SCRD28 , n=56, 59 | 0.989 [0.722 to 1.355] | 1.220 [0.909 to 1.637]
  TLC; Scan Trimmed; Lobes; RML; D12D28 , n =56, 58 | 1.102 [0.869 to 1.397] | 0.988 [0.771 to 1.266]
  TLC; Scan Trimmed; Lobes; RLL; SCRD12 , n =56, 59 | 0.848 [0.587 to 1.225] | 1.143 [0.900 to 1.451]
  TLC; Scan Trimmed; Lobes; RLL; SCRD28 , n=56, 58 | 0.965 [0.688 to 1.352] | 1.122 [0.868 to 1.452]
  TLC; Scan Trimmed; Lobes; RLL; D12D28 , n =53, 57 | 1.208 [0.941 to 1.550] | 0.927 [0.775 to 1.109]
  TLC; Scan Trimmed; Lobes; LLL; SCRD12 , n =55, 59 | 0.813 [0.605 to 1.093] | 1.139 [0.893 to 1.453]
  TLC; Scan Trimmed; Lobes; LLL; SCRD28 , n=55, 58 | 0.958 [0.682 to 1.346] | 0.987 [0.758 to 1.285]
  TLC; Scan Trimmed; Lobes; LLL; D12D28 , n=52, 57 | 1.313 [1.022 to 1.686] | 0.829 [0.670 to 1.026]
  TLC; Scan Trimmed; Region;Upper; SCRD12 ,n =56, 59 | 0.913 [0.754 to 1.106] | 1.103 [0.911 to 1.335]
  TLC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 58 | 0.958 [0.751 to 1.222] | 0.957 [0.764 to 1.200]
  TLC; Scan Trimmed; Region;Upper; D12D28 ,n =53, 57 | 1.067 [0.896 to 1.270] | 0.885 [0.752 to 1.040]
  TLC; Scan Trimmed; Region;Lower; SCRD12 ,n =56, 59 | 0.850 [0.621 to 1.163] | 1.116 [0.897 to 1.388]
  TLC; Scan Trimmed; Region; Lower; SCRD28 ,n=56, 58 | 0.953 [0.676 to 1.344] | 1.056 [0.827 to 1.347]
  TLC; Scan Trimmed; Region;Lower; D12D28 ,n =53, 57 | 1.269 [1.021 to 1.578] | 0.862 [0.723 to 1.028]
  TLC;Scan Trimmed;Region;Central; SCRD12 ,n =56, 59 | 0.960 [0.841 to 1.095] | 1.007 [0.937 to 1.081]
  TLC;Scan Trimmed; Region Central; SCRD28 ,n=56, 58 | 0.976 [0.838 to 1.136] | 1.000 [0.933 to 1.070]
  TLC;Scan Trimmed;Region Central; D12D28 ,n =53, 57 | 1.039 [0.945 to 1.142] | 0.981 [0.932 to 1.032]
  TLC;Scan Trimmed; Region;Distal; SCRD12 ,n =56, 59 | 0.889 [0.680 to 1.161] | 1.116 [0.913 to 1.364]
  TLC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 58 | 0.945 [0.698 to 1.279] | 0.976 [0.793 to 1.201]
  TLC;Scan Trimmed;Region;Distal; D12D28 , n =53, 57 | 1.189 [1.000 to 1.414] | 0.838 [0.719 to 0.976]
  TLC;Scan Trimmed; Region;Total; SCRD12 , n =56, 59 | 0.891 [0.762 to 1.042] | 1.061 [0.937 to 1.202]
  TLC;Scan Trimmed;Region;Total; SCRD28 , n=56, 58 | 0.956 [0.781 to 1.171] | 0.989 [0.861 to 1.136]
  TLC; Scan Trimmed;Region;Total; D12D28 , n =53, 57 | 1.133 [0.990 to 1.296] | 0.904 [0.816 to 1.002]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 60.07, Bayesian repeated measures model — The data entered for the p-value represents the posterior probability that the true treatment ratio is less than 1. P-value is denoted in percentage; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.66 to 1.39] — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 51.75, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.65 to 1.53] — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 65.66, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.60 to 1.40] — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 81.67, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.85, 95% CI 2-sided [0.59 to 1.21] — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 5: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 89.98, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.77, 95% CI 2-sided [0.51 to 1.15] — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 6: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 43.88, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.70 to 1.51] — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 7: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 36.10, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.10, 95% CI 2-sided [0.64 to 1.91] — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 8: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.74, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.70, 95% CI 2-sided [0.47 to 1.05] — [estimate comment as in outcome 1, analysis 18]
Statistical Analysis 9: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 50.74, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.67 to 1.48] — [estimate comment as in outcome 1, analysis 19]
Statistical Analysis 10: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 72.81, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.85, 95% CI 2-sided [0.51 to 1.44] — [estimate comment as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.41, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.73, 95% CI 2-sided [0.50 to 1.08] — [estimate comment as in outcome 1, analysis 21]
Statistical Analysis 12: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 81.07, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.83, 95% CI 2-sided [0.55 to 1.25] — [estimate comment as in outcome 1, analysis 22]
Statistical Analysis 13: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 69.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.87, 95% CI 2-sided [0.50 to 1.51] — [estimate comment as in outcome 1, analysis 23]
Statistical Analysis 14: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 73.67, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.86, 95% CI 2-sided [0.54 to 1.37] — [estimate comment as in outcome 1, analysis 24]
Statistical Analysis 15: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.82, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.87, 95% CI 2-sided [0.59 to 1.29] — [estimate comment as in outcome 1, analysis 25]
Statistical Analysis 16: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 54.22, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.69 to 1.39] — FRC; Scan Trimmed; Region; Upper; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 17: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 66.46, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.63 to 1.35] — FRC; Scan Trimmed; Region; Upper; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 18: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 21.45, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.16, 95% CI 2-sided [0.79 to 1.71] — FRC; Scan Trimmed; Region; Upper; D12D28 . The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 19: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 69.91, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.86, 95% CI 2-sided [0.50 to 1.50] — FRC; Scan Trimmed; Region; Lower; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 20: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.86, 95% CI 2-sided [0.57 to 1.31] — [estimate comment as in outcome 1, analysis 40]
Statistical Analysis 21: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 44.05, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.68 to 1.58] — FRC; Scan Trimmed; Region; Lower; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 22: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.93, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.82, 95% CI 2-sided [0.65 to 1.04] — FRC;Scan Trimmed; Region; Central; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 23: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.11, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.77, 95% CI 2-sided [0.59 to 1.01] — FRC; Scan Trimmed; Region Central; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 24: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 85.41, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.70 to 1.11] — FRC; Scan Trimmed; Region Central; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 25: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 54.73, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.62 to 1.53] — FRC; Scan Trimmed; Region; Distal; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 26: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 72.31, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.61 to 1.30] — FRC; Scan Trimmed; Region; Distal; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 27: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 15.05, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.21, 95% CI 2-sided [0.84 to 1.75] — FRC; Scan Trimmed; Region; Distal; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 28: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 84.87, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.88, 95% CI 2-sided [0.68 to 1.13] — FRC; Scan Trimmed; Region; Total; SCRD12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 29: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 92.24, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.82, 95% CI 2-sided [0.63 to 1.08] — FRC; Scan Trimmed; Region; Total; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 30: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.42, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.75 to 1.22] — FRC; Scan Trimmed; Region; Total; D12D28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 31: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.05, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.17, 95% CI 2-sided [0.93 to 1.46] — [estimate comment as in outcome 1, analysis 61]
Statistical Analysis 32: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 66.40, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.74 to 1.22] — [estimate comment as in outcome 1, analysis 62]
Statistical Analysis 33: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 97.39, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.78, 95% CI 2-sided [0.60 to 1.00] — [estimate comment as in outcome 1, analysis 63]
Statistical Analysis 34: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 16.02, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.13, 95% CI 2-sided [0.89 to 1.42] — [estimate comment as in outcome 1, analysis 64]
Statistical Analysis 35: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.69, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.90, 95% CI 2-sided [0.68 to 1.21] — [estimate comment as in outcome 1, analysis 65]
Statistical Analysis 36: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 90.22, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.86, 95% CI 2-sided [0.69 to 1.08] — [estimate comment as in outcome 1, analysis 66]
Statistical Analysis 37: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.64, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.21, 95% CI 2-sided [0.91 to 1.62] — [estimate comment as in outcome 1, analysis 67]
Statistical Analysis 38: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 20.44, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.15, 95% CI 2-sided [0.82 to 1.61] — [estimate comment as in outcome 1, analysis 68]
Statistical Analysis 39: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 55.06, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.73 to 1.31] — [estimate comment as in outcome 1, analysis 69]
Statistical Analysis 40: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 5.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.36, 95% CI 2-sided [0.94 to 1.97] — [estimate comment as in outcome 1, analysis 70]
Statistical Analysis 41: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 28.82, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.11, 95% CI 2-sided [0.77 to 1.60] — [estimate comment as in outcome 1, analysis 71]
Statistical Analysis 42: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 93.00, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.81, 95% CI 2-sided [0.61 to 1.07] — [estimate comment as in outcome 1, analysis 72]
Statistical Analysis 43: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 1.64, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.42, 95% CI 2-sided [1.03 to 1.95] — [estimate comment as in outcome 1, analysis 73]
Statistical Analysis 44: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 50.71, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.72 to 1.38] — [estimate comment as in outcome 1, analysis 74]
Statistical Analysis 45: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.52, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.68, 95% CI 2-sided [0.51 to 0.91] — [estimate comment as in outcome 1, analysis 75]
Statistical Analysis 46: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 3.10, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.22, 95% CI 2-sided [0.99 to 1.51] — [estimate comment as in outcome 2, analysis 86]
Statistical Analysis 47: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.39, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.71 to 1.18] — [estimate comment as in outcome 2, analysis 87]
Statistical Analysis 48: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 93.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.85, 95% CI 2-sided [0.68 to 1.05] — [estimate comment as in outcome 2, analysis 88]
Statistical Analysis 49: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 3.79, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.33, 95% CI 2-sided [0.97 to 1.82] — [estimate comment as in outcome 1, analysis 89]
Statistical Analysis 50: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 36.75, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.76 to 1.48] — [estimate comment as in outcome 1, analysis 90]
Statistical Analysis 51: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.32, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.72, 95% CI 2-sided [0.56 to 0.93] — [estimate comment as in outcome 1, analysis 91]
Statistical Analysis 52: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 18.91, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.06, 95% CI 2-sided [0.93 to 1.20] — [estimate comment as in outcome 1, analysis 92]
Statistical Analysis 53: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 47.35, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.87 to 1.15] — [estimate comment as in outcome 1, analysis 93]
Statistical Analysis 54: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 78.00, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.96, 95% CI 2-sided [0.86 to 1.07] — [estimate comment as in outcome 1, analysis 94]
Statistical Analysis 55: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 2.65, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.29, 95% CI 2-sided [1.00 to 1.67] — [estimate comment as in outcome 1, analysis 95]
Statistical Analysis 56: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 58.48, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.73 to 1.29] — [estimate comment as in outcome 1, analysis 96]
Statistical Analysis 57: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.64, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 21]; Posterior Median Ratio = 0.75, 95% CI 2-sided [0.61 to 0.92] — [estimate comment as in outcome 1, analysis 97]
Statistical Analysis 58: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 1.90, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.19, 95% CI 2-sided [1.01 to 1.40] — [estimate comment as in outcome 1, analysis 98]
Statistical Analysis 59: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.03, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.97, 95% CI 2-sided [0.81 to 1.16] — [estimate comment as in outcome 1, analysis 99]
Statistical Analysis 60: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.19, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.83, 95% CI 2-sided [0.72 to 0.97] — [estimate comment as in outcome 1, analysis 100]

4. Secondary Outcome: Change From Baseline in Imaging Specific Airways Resistance: siRaw Measured at FRC and TLC Scan Conditions, Presented in Scan Trimmed Scan Types, Measured in 5 Lobes and 5 Regions at Screening, Day 12 and Day 28
Description: siRaw was derived from HRCT to evaluate the effect of once daily inhaled dose of GSK2269557 on lung parameters. It was measured at functional residual volume (FRC) and total lung capacity (TLC). Data was collected at each time point for scan trimmed pairs: SCRD12, SCRD28 & D12D28. At each time point it was measure at 5 lobes (RUL, LUL, RML, RLL & LLL) and 5 Regions (Upper, Lower, Central, Distal & Total). For SCRD12 & SCRD28 scan trimmed pairs the baseline is screening, for D12D28 scan trimmed pair the baseline is D12. Change from baseline is the post-Baseline value minus the Baseline value. Only particpants available at the specified time point were analysed (represented by n=X1, X2 in the category title).
Time Frame: Baseline, Day 12 and Day 28
Population: ITT Population excluding the subject with a pacemaker.
Measure: Geometric Mean (95% Confidence Interval); unit: Kpa*s
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 62 | 63
Kpa*s
  FRC; Scan Trimmed; Lobes; RUL; SCRD12 , n =54, 57 | 0.896 [0.613 to 1.310] | 0.908 [0.669 to 1.231]
  FRC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 56 | 0.829 [0.516 to 1.333] | 1.013 [0.757 to 1.355]
  FRC; Scan Trimmed; Lobes; RUL; D12D28 , n =51, 55 | 1.035 [0.712 to 1.505] | 0.926 [0.720 to 1.191]
  FRC; Scan Trimmed; Lobes; LUL; SCRD12 , n =56, 59 | 0.957 [0.671 to 1.365] | 0.944 [0.715 to 1.247]
  FRC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 58 | 0.919 [0.610 to 1.383] | 0.834 [0.585 to 1.189]
  FRC; Scan Trimmed; Lobes; LUL; D12D28 , n =53, 57 | 0.849 [0.608 to 1.184] | 0.948 [0.717 to 1.254]
  FRC; Scan Trimmed; Lobes; RML; SCRD12 , n =52, 58 | 1.009 [0.655 to 1.553] | 1.013 [0.669 to 1.533]
  FRC; Scan Trimmed; Lobes; RML; SCRD28 , n=53, 57 | 1.349 [0.856 to 2.125] | 0.904 [0.649 to 1.261]
  FRC; Scan Trimmed; Lobes; RML; D12D28 , n =52, 56 | 1.028 [0.695 to 1.521] | 1.213 [0.818 to 1.798]
  FRC; Scan Trimmed; Lobes; RLL; SCRD12 , n =54, 59 | 1.078 [0.687 to 1.691] | 1.046 [0.671 to 1.632]
  FRC; Scan Trimmed; Lobes; RLL; SCRD28 , n=55, 58 | 1.468 [0.990 to 2.177] | 1.053 [0.736 to 1.507]
  FRC; Scan Trimmed; Lobes; RLL; D12D28 , n =52, 57 | 1.284 [0.940 to 1.754] | 1.130 [0.778 to 1.641]
  FRC; Scan Trimmed; Lobes; LLL; SCRD12 , n =53, 58 | 0.755 [0.506 to 1.127] | 0.725 [0.479 to 1.098]
  FRC; Scan Trimmed; Lobes; LLL; SCRD28 , n=54, 58 | 0.930 [0.629 to 1.375] | 0.811 [0.539 to 1.220]
  FRC; Scan Trimmed; Lobes; LLL; D12D28 , n =51, 56 | 1.063 [0.829 to 1.362] | 1.017 [0.702 to 1.476]
  FRC; Scan Trimmed; Region;Upper; SCRD12 ,n =56, 59 | 0.915 [0.645 to 1.300] | 0.956 [0.740 to 1.237]
  FRC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 58 | 0.919 [0.617 to 1.370] | 0.898 [0.659 to 1.223]
  FRC; Scan Trimmed; Region;Upper; D12D28 ,n =53, 57 | 0.870 [0.620 to 1.220] | 1.142 [0.849 to 1.536]
  FRC; Scan Trimmed; Region;Lower; SCRD12 ,n =54, 59 | 0.825 [0.530 to 1.283] | 0.816 [0.524 to 1.270]
  FRC; Scan Trimmed; Region; Lower; SCRD28 ,n=55, 58 | 1.188 [0.821 to 1.718] | 0.869 [0.606 to 1.246]
  FRC; Scan Trimmed; Region;Lower; D12D28 ,n =52, 57 | 1.114 [0.881 to 1.409] | 1.200 [0.810 to 1.777]
  FRC;Scan Trimmed;Region;Central; SCRD12 ,n =56, 59 | 1.077 [0.813 to 1.425] | 0.928 [0.762 to 1.130]
  FRC;Scan Trimmed; Region Central; SCRD28 ,n=56, 58 | 1.053 [0.777 to 1.427] | 0.957 [0.817 to 1.121]
  FRC;Scan Trimmed;Region Central; D12D28 ,n =53, 57 | 1.035 [0.851 to 1.259] | 1.022 [0.863 to 1.210]
  FRC;Scan Trimmed; Region;Distal; SCRD12 ,n =56, 59 | 0.781 [0.533 to 1.144] | 0.854 [0.598 to 1.220]
  FRC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 58 | 0.969 [0.661 to 1.421] | 0.880 [0.645 to 1.202]
  FRC;Scan Trimmed;Region;Distal; D12D28 , n =53, 57 | 0.890 [0.672 to 1.179] | 1.234 [0.903 to 1.687]
  FRC;Scan Trimmed; Region;Total; SCRD12 , n =56, 59 | 0.982 [0.741 to 1.300] | 0.914 [0.732 to 1.140]
  FRC;Scan Trimmed;Region;Total; SCRD28 , n=56, 58 | 1.012 [0.742 to 1.378] | 0.929 [0.760 to 1.136]
  FRC; Scan Trimmed;Region;Total; D12D28 , n =53, 57 | 1.003 [0.821 to 1.225] | 1.078 [0.886 to 1.311]
  TLC; Scan Trimmed; Lobes; RUL; SCRD12 , n =56, 59 | 0.848 [0.686 to 1.049] | 0.989 [0.816 to 1.198]
  TLC; Scan Trimmed; Lobes; RUL; SCRD28 , n=56, 58 | 0.934 [0.725 to 1.203] | 1.043 [0.846 to 1.285]
  TLC; Scan Trimmed; Lobes; RUL; D12D28 , n =53, 57 | 1.142 [0.945 to 1.379] | 0.903 [0.757 to 1.077]
  TLC; Scan Trimmed; Lobes; LUL; SCRD12 , n =56, 59 | 0.880 [0.721 to 1.074] | 0.977 [0.832 to 1.148]
  TLC; Scan Trimmed; Lobes; LUL; SCRD28 , n=56, 58 | 0.926 [0.736 to 1.165] | 0.885 [0.690 to 1.134]
  TLC; Scan Trimmed; Lobes; LUL; D12D28 , n =53, 57 | 1.023 [0.856 to 1.221] | 0.896 [0.751 to 1.069]
  TLC; Scan Trimmed; Lobes; RML; SCRD12 , n =57, 58 | 1.073 [0.829 to 1.390] | 1.343 [0.995 to 1.814]
  TLC; Scan Trimmed; Lobes; RML; SCRD28 , n=56, 59 | 0.981 [0.727 to 1.324] | 1.238 [0.921 to 1.664]
  TLC; Scan Trimmed; Lobes; RML; D12D28 , n =56, 58 | 1.093 [0.867 to 1.377] | 1.010 [0.782 to 1.303]
  TLC; Scan Trimmed; Lobes; RLL; SCRD12 , n =56, 59 | 0.854 [0.595 to 1.226] | 1.149 [0.910 to 1.449]
  TLC; Scan Trimmed; Lobes; RLL; SCRD28 , n=56, 58 | 0.964 [0.695 to 1.337] | 1.134 [0.887 to 1.450]
  TLC; Scan Trimmed; Lobes; RLL; D12D28 , n =53, 57 | 1.192 [0.937 to 1.518] | 0.935 [0.782 to 1.117]
  TLC; Scan Trimmed; Lobes; LLL; SCRD12 , n =55, 59 | 0.820 [0.617 to 1.089] | 1.126 [0.891 to 1.424]
  TLC; Scan Trimmed; Lobes; LLL; SCRD28 , n=55, 58 | 0.960 [0.690 to 1.335] | 0.985 [0.760 to 1.276]
  TLC; Scan Trimmed; Lobes; LLL; D12D28 , n=52, 57 | 1.302 [1.013 to 1.674] | 0.839 [0.679 to 1.037]
  TLC; Scan Trimmed; Region;Upper; SCRD12 ,n =56, 59 | 0.917 [0.760 to 1.106] | 1.100 [0.912 to 1.327]
  TLC; Scan Trimmed; Region;Upper; SCRD28 ,n=56, 58 | 0.961 [0.762 to 1.213] | 0.957 [0.767 to 1.195]
  TLC; Scan Trimmed; Region;Upper; D12D28 ,n =53, 57 | 1.060 [0.891 to 1.262] | 0.888 [0.755 to 1.045]
  TLC; Scan Trimmed; Region;Lower; SCRD12 ,n =56, 59 | 0.856 [0.631 to 1.162] | 1.112 [0.900 to 1.374]
  TLC; Scan Trimmed; Region; Lower; SCRD28 ,n=56, 58 | 0.954 [0.683 to 1.332] | 1.061 [0.838 to 1.342]
  TLC; Scan Trimmed; Region;Lower; D12D28 ,n =53, 57 | 1.256 [1.015 to 1.553] | 0.871 [0.731 to 1.038]
  TLC;Scan Trimmed;Region;Central; SCRD12 ,n =56, 59 | 0.963 [0.850 to 1.092] | 1.004 [0.931 to 1.083]
  TLC;Scan Trimmed; Region Central; SCRD28 ,n=56, 58 | 0.977 [0.852 to 1.121] | 1.002 [0.927 to 1.082]
  TLC;Scan Trimmed;Region Central; D12D28 ,n =53, 57 | 1.032 [0.939 to 1.135] | 0.988 [0.941 to 1.037]
  TLC;Scan Trimmed; Region;Distal; SCRD12 ,n =56, 59 | 0.892 [0.688 to 1.157] | 1.112 [0.915 to 1.353]
  TLC;Scan Trimmed;Region; Distal; SCRD28 , n=56, 58 | 0.946 [0.705 to 1.270] | 0.978 [0.800 to 1.195]
  TLC;Scan Trimmed;Region;Distal; D12D28 , n =53, 57 | 1.181 [0.996 to 1.401] | 0.844 [0.724 to 0.983]
  TLC;Scan Trimmed; Region;Total; SCRD12 , n =56, 59 | 0.895 [0.771 to 1.038] | 1.058 [0.938 to 1.194]
  TLC;Scan Trimmed;Region;Total; SCRD28 , n=56, 58 | 0.958 [0.793 to 1.158] | 0.991 [0.867 to 1.133]
  TLC; Scan Trimmed;Region;Total; D12D28 , n =53, 57 | 1.125 [0.986 to 1.285] | 0.911 [0.822 to 1.008]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 67.19, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.64 to 1.33] — [estimate comment as in outcome 1, analysis 11]
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 44.80, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.66 to 1.61] — [estimate comment as in outcome 1, analysis 12]
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 59.90, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.61 to 1.46] — [estimate comment as in outcome 1, analysis 13]
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 70.12, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.91, 95% CI 2-sided [0.63 to 1.31] — [estimate comment as in outcome 1, analysis 14]
Statistical Analysis 5: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 83.98, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.82, 95% CI 2-sided [0.54 to 1.22] — [estimate comment as in outcome 1, analysis 15]
Statistical Analysis 6: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 34.93, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.08, 95% CI 2-sided [0.73 to 1.57] — [estimate comment as in outcome 1, analysis 16]
Statistical Analysis 7: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 32.45, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.14, 95% CI 2-sided [0.65 to 1.96] — [estimate comment as in outcome 1, analysis 17]
Statistical Analysis 8: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 95.35, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.70, 95% CI 2-sided [0.46 to 1.06] — [estimate comment as in outcome 1, analysis 18]
Statistical Analysis 9: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 50.10, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.66 to 1.54] — [estimate comment as in outcome 1, analysis 19]
Statistical Analysis 10: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 59.37, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.94, 95% CI 2-sided [0.55 to 1.60] — [estimate comment as in outcome 1, analysis 20]
Statistical Analysis 11: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 87.99, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.80, 95% CI 2-sided [0.55 to 1.17] — [estimate comment as in outcome 1, analysis 21]
Statistical Analysis 12: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 70.87, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.59 to 1.36] — [estimate comment as in outcome 1, analysis 22]
Statistical Analysis 13: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.71, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.91, 95% CI 2-sided [0.51 to 1.60] — [estimate comment as in outcome 1, analysis 23]
Statistical Analysis 14: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 65.99, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.91, 95% CI 2-sided [0.57 to 1.44] — [estimate comment as in outcome 1, analysis 24]
Statistical Analysis 15: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 71.95, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.89, 95% CI 2-sided [0.60 to 1.32] — [estimate comment as in outcome 1, analysis 25]
Statistical Analysis 16: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 48.28, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.71 to 1.43] — [estimate comment as in outcome 1, analysis 36]
Statistical Analysis 17: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 61.06, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.95, 95% CI 2-sided [0.65 to 1.39] — [estimate comment as in outcome 1, analysis 37]
Statistical Analysis 18: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 18.05, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.19, 95% CI 2-sided [0.82 to 1.74] — [estimate comment as in outcome 1, analysis 38]
Statistical Analysis 19: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 61.12, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.53 to 1.61] — [estimate comment as in outcome 1, analysis 39]
Statistical Analysis 20: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 64.40, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.92, 95% CI 2-sided [0.61 to 1.41] — [estimate comment as in outcome 1, analysis 40]
Statistical Analysis 21: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 38.12, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.69 to 1.66] — [estimate comment as in outcome 1, analysis 41]
Statistical Analysis 22: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 91.00, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.85, 95% CI 2-sided [0.67 to 1.08] — [estimate comment as in outcome 1, analysis 42]
Statistical Analysis 23: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 94.52, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.81, 95% CI 2-sided [0.62 to 1.05] — [estimate comment as in outcome 1, analysis 43]
Statistical Analysis 24: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 82.11, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.90, 95% CI 2-sided [0.72 to 1.13] — [estimate comment as in outcome 1, analysis 44]
Statistical Analysis 25: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 48.10, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.64 to 1.60] — [estimate comment as in outcome 1, analysis 45]
Statistical Analysis 26: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 65.66, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.93, 95% CI 2-sided [0.64 to 1.36] — [estimate comment as in outcome 2, analysis 46]
Statistical Analysis 27: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 11.46, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.25, 95% CI 2-sided [0.87 to 1.80] — [estimate comment as in outcome 1, analysis 47]
Statistical Analysis 28: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 77.20, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.91, 95% CI 2-sided [0.70 to 1.17] — [estimate comment as in outcome 1, analysis 48]
Statistical Analysis 29: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 87.35, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.86, 95% CI 2-sided [0.66 to 1.11] — [estimate comment as in outcome 1, analysis 49]
Statistical Analysis 30: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 56.53, Bayesian repeated measures random effect — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.77 to 1.25] — [estimate comment as in outcome 1, analysis 50]
Statistical Analysis 31: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 7.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.19, 95% CI 2-sided [0.94 to 1.50] — [estimate comment as in outcome 1, analysis 61]
Statistical Analysis 32: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 55.09, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.75 to 1.28] — [estimate comment as in outcome 1, analysis 62]
Statistical Analysis 33: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 96.49, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.79, 95% CI 2-sided [0.61 to 1.02] — [estimate comment as in outcome 1, analysis 63]
Statistical Analysis 34: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 14.54, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.13, 95% CI 2-sided [0.90 to 1.44] — [estimate comment as in outcome 1, analysis 64]
Statistical Analysis 35: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 66.85, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.94, 95% CI 2-sided [0.71 to 1.25] — [estimate comment as in outcome 1, analysis 65]
Statistical Analysis 36: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 85.77, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.88, 95% CI 2-sided [0.70 to 1.11] — [estimate comment as in outcome 1, analysis 66]
Statistical Analysis 37: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 8.67, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.24, 95% CI 2-sided [0.91 to 1.70] — [estimate comment as in outcome 1, analysis 67]
Statistical Analysis 38: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 14.80, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.22, 95% CI 2-sided [0.84 to 1.75] — [estimate comment as in outcome 1, analysis 68]
Statistical Analysis 39: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 45.69, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.75 to 1.37] — [estimate comment as in outcome 1, analysis 69]
Statistical Analysis 40: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 2.94, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.42, 95% CI 2-sided [0.99 to 2.06] — [estimate comment as in outcome 1, analysis 70]
Statistical Analysis 41: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 13.92, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.22, 95% CI 2-sided [0.85 to 1.73] — [estimate comment as in outcome 1, analysis 71]
Statistical Analysis 42: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 86.40, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.86, 95% CI 2-sided [0.65 to 1.13] — [estimate comment as in outcome 1, analysis 72]
Statistical Analysis 43: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.88, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.46, 95% CI 2-sided [1.06 to 2.00] — [estimate comment as in outcome 1, analysis 73]
Statistical Analysis 44: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 41.25, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.75 to 1.43] — [estimate comment as in outcome 1, analysis 74]
Statistical Analysis 45: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.20, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.70, 95% CI 2-sided [0.52 to 0.94] — [estimate comment as in outcome 1, analysis 75]
Statistical Analysis 46: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 3.49, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.22, 95% CI 2-sided [0.98 to 1.51] — TLC; Scan Trimmed; Region;Upper; SCRD12 .The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 47: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 73.09, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.93, 95% CI 2-sided [0.72 to 1.19] — TLC; Scan Trimmed; Region;Upper; SCRD28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 48: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 92.41, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.85, 95% CI 2-sided [0.69 to 1.06] — [estimate comment as in outcome 1, analysis 88]
Statistical Analysis 49: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 2.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.38, 95% CI 2-sided [1.01 to 1.89] — [estimate comment as in outcome 1, analysis 89]
Statistical Analysis 50: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 23.67, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; Non-informative priors used for all modelling parameters.Unstructured covariance matrix fitted, accounting for correlation within region and visit; Posterior Median Ratio = 1.12, 95% CI 2-sided [0.81 to 1.56] — [estimate comment as in outcome 1, analysis 90]
Statistical Analysis 51: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.87, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.75, 95% CI 2-sided [0.59 to 0.96] — [estimate comment as in outcome 1, analysis 91]
Statistical Analysis 52: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 14.50, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.07, 95% CI 2-sided [0.95 to 1.20] — [estimate comment as in outcome 1, analysis 92]
Statistical Analysis 53: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 30.26, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.91 to 1.18] — [estimate comment as in outcome 1, analysis 93]
Statistical Analysis 54: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 62.84, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.89 to 1.09] — TLC;Scan Trimmed;Region Central; D12D28 .The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 55: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 2.06, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.31, 95% CI 2-sided [1.01 to 1.70] — [estimate comment as in outcome 1, analysis 95]
Statistical Analysis 56: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 49.97, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.76 to 1.32] — [estimate comment as in outcome 1, analysis 96]
Statistical Analysis 57: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 99.43, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.76, 95% CI 2-sided [0.62 to 0.94] — [estimate comment as in outcome 1, analysis 97]
Statistical Analysis 58: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 1.17, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.20, 95% CI 2-sided [1.02 to 1.41] — [estimate comment as in outcome 1, analysis 98]
Statistical Analysis 59: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 49.78, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.84 to 1.18] — [estimate comment as in outcome 1, analysis 99]
Statistical Analysis 60: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 98.66, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.85, 95% CI 2-sided [0.73 to 0.98] — [estimate comment as in outcome 1, analysis 100]

5. Secondary Outcome: Change From Baseline in Lung Lobar Volumes Measured at FRC and TLC Scan Conditions, Presented in Longitudinal Scan Types, Measured in 5 Lobes and 5 Regions at Day 12 and Day 28
Description: Change from Baseline in lung lobar volumes was measured at functional residual volume (FRC) and total lung capacity (TLC) scan conditions. Data was collected at longitudinal time points: Day 12 & Day 28. At each time point it was measure at 5 lobes (RUL, LUL, RML, RLL & LLL) and 5 Regions (Upper, Lower, Central, Distal & Total). For longitudinal time points the baseline is screening. Change from baseline is the post-Baseline value minus the Baseline value. Only particpants available at the specified time point were analysed (represented by n=X1, X2 in the category title).
Time Frame: Baseline, Day 12 and Day 28
Population: ITT Population excluding the subject with a pacemaker.
Measure: Geometric Mean (95% Confidence Interval); unit: L
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 62 | 63
L
  FRC Lobes; RUL; Day 12, n =56, 57 | 0.983 [0.953 to 1.014] | 0.995 [0.964 to 1.026]
  FRC Lobes; RUL Day 28, n =56, 56 | 0.977 [0.949 to 1.005] | 1.017 [0.985 to 1.050]
  FRC Lobes; LUL Day 12, n =56, 59 | 0.974 [0.943 to 1.007] | 0.998 [0.964 to 1.034]
  FRC Lobes;LUL Day 28, n =56, 58 | 0.980 [0.953 to 1.009] | 1.017 [0.978 to 1.057]
  FRC Lobes; RML Day 12, n =55, 58 | 0.981 [0.943 to 1.022] | 0.992 [0.959 to 1.025]
  FRC Lobes; RML Day 28, n =56, 57 | 0.972 [0.943 to 1.002] | 0.996 [0.963 to 1.030]
  FRC Lobes; RLL Day 12, n =56, 59 | 0.977 [0.933 to 1.024] | 1.004 [0.964 to 1.045]
  FRC Lobes; RLL Day 28, n =56, 58 | 0.972 [0.939 to 1.007] | 1.009 [0.968 to 1.051]
  FRC Lobes; LLL Day 12, n =55, 59 | 0.968 [0.934 to 1.004] | 0.983 [0.944 to 1.024]
  FRC Lobes; LLL Day 28, n =55, 58 | 0.979 [0.948 to 1.010] | 0.991 [0.950 to 1.033]
  FRC Region; Upper Day 12, n =56, 59 | 0.980 [0.950 to 1.011] | 0.996 [0.966 to 1.027]
  FRC Region; Upper Day 28, n =56, 58 | 0.978 [0.954 to 1.004] | 1.013 [0.979 to 1.047]
  FRC Region; Lower Day 12, n =56, 59 | 0.975 [0.936 to 1.016] | 0.994 [0.956 to 1.033]
  FRC Region; Lower Day 28, n =56, 58 | 0.975 [0.945 to 1.007] | 1.001 [0.962 to 1.041]
  FRC Region; Total Day 12, n =56, 59 | 0.975 [0.944 to 1.007] | 0.994 [0.964 to 1.026]
  FRC Region; Total Day 28, n =56, 58 | 0.976 [0.950 to 1.003] | 1.008 [0.974 to 1.042]
  TLC Lobes; RUL; Day 12, n =58, 57 | 1.009 [0.994 to 1.024] | 0.999 [0.986 to 1.011]
  TLC Lobes; RUL Day 28, n =56, 57 | 1.005 [0.985 to 1.025] | 0.999 [0.984 to 1.013]
  TLC Lobes; LUL Day 12, n =58, 59 | 1.002 [0.989 to 1.014] | 0.998 [0.984 to 1.013]
  TLC Lobes;LUL Day 28, n =56, 59 | 1.004 [0.984 to 1.025] | 0.998 [0.982 to 1.014]
  TLC Lobes; RML Day 12, n =57, 58 | 0.998 [0.975 to 1.021] | 0.988 [0.970 to 1.005]
  TLC Lobes; RML Day 28, n =56, 58 | 0.992 [0.960 to 1.025] | 0.996 [0.979 to 1.013]
  TLC Lobes; RLL Day 12, n =58, 59 | 1.010 [0.983 to 1.038] | 1.005 [0.977 to 1.034]
  TLC Lobes; RLL Day 28, n =56, 59 | 1.000 [0.974 to 1.026] | 1.009 [0.975 to 1.044]
  TLC Lobes; LLL Day 12, n =57, 59 | 1.008 [0.975 to 1.042] | 0.989 [0.964 to 1.014]
  TLC Lobes; LLL Day 28, n =55, 59 | 1.002 [0.977 to 1.028] | 0.996 [0.968 to 1.024]
  TLC Upper Day 12, n =58, 59 | 1.005 [0.993 to 1.017] | 0.997 [0.985 to 1.010]
  TLC UpperDay 28, n =56, 59 | 1.004 [0.984 to 1.023] | 0.999 [0.985 to 1.012]
  TLC Lower Day 12, n =58, 59 | 1.009 [0.982 to 1.037] | 0.997 [0.972 to 1.023]
  TLC Lower Day 28, n =56, 59 | 1.000 [0.978 to 1.024] | 1.003 [0.973 to 1.034]
  TLC Total Day 12, n =58, 59 | 1.005 [0.989 to 1.022] | 0.997 [0.980 to 1.015]
  TLC Total Day 28, n =56, 59 | 1.002 [0.982 to 1.022] | 1.001 [0.981 to 1.021]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 32.51, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.97 to 1.06] — FRC Lobes; RUL; Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 6.21, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.99 to 1.08] — FRC Lobes; RUL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 15.91, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.98 to 1.07] — FRC Lobes; LUL Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 6.73, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.99 to 1.09] — FRC Lobes;LUL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 5: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 27.65, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.96 to 1.07] — FRC Lobes; RML Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 6: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 12.19, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.98 to 1.07] — FRC Lobes; RML Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 7: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 11.62, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.98 to 1.10] — FRC Lobes; RLL Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 8: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 7.66, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [0.99 to 1.10] — FRC Lobes; RLL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 9: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 28.88, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.96 to 1.07] — FRC Lobes; LLL Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 10: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 28.28, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.96 to 1.07] — FRC Lobes; LLL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 11: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 27.87, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.97 to 1.05] — FRC Region; Upper Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 12: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 9.83, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 21]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.99 to 1.07] — FRC Region; Upper Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 13: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 21.87, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.97 to 1.07] — FRC Region; Lower Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 14: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 18.58, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.97 to 1.07] — FRC Region; Lower Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 15: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 22.28, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.98 to 1.06] — FRC Region; Total Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 16: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 10.86, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.03, 95% CI 2-sided [0.98 to 1.07] — FRC Region; Total Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 17: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 84.89, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.97 to 1.01] — TLC Lobes; RUL; Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 18: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.78, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.97 to 1.02] — TLC Lobes; RUL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 19: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 69.42, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.98 to 1.01] — TLC Lobes; LUL Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 20: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 62.63, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.97 to 1.02] — TLC Lobes;LUL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 21: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 72.55, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.02] — TLC Lobes; RML Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 22: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 36.28, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.97 to 1.04] — TLC Lobes; RML Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 23: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 47.44, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.96 to 1.04] — TLC Lobes; RLL Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 24: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 22.99, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.97 to 1.06] — TLC Lobes; RLL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 25: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 85.95, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.98, 95% CI 2-sided [0.94 to 1.02] — TLC Lobes; LLL Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 26: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 60.20, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.03] — TLC Lobes; LLL Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 27: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 81.34, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.97 to 1.01] — TLC Upper Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 28: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 63.04, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.97 to 1.02] — TLC UpperDay 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 29: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 69.67, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.96 to 1.03] — TLC Lower Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 30: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 39.81, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.97 to 1.04] — TLC Lower Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 31: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 73.01, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.97 to 1.02] — TLC Total Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 32: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 48.97, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.97 to 1.03] — TLC Total Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval

6. Secondary Outcome: Change From Baseline in Imaging Trachea Length and Diameter After 12 Days of Treatment and After 28 Days of Treatment
Description: Imaging trachea length and diameter was derived from HRCT to evaluate the effect of once daily inhaled dose of GSK2269557 on lung parameters. TLC is the volume in the lungs at maximal inflation and FRC is the volume in the lungs at the end-expiratory position. The Baseline for the assessment on Day 12 and Day 28 is the Screening value. Change from Baseline is the post-Baseline value minus the Baseline value. The change from Baseline data is presented for Day 12 and Day 28 for trachea length and diameter. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 12 and Day 28
Population: ITT Population excluding the subject with a pacemaker.
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 62 | 63
Millimeter (mm)
  FRC Length Day 12, n=56, 59 | -1.886 (7.6043) | 0.517 (6.0882)
  FRC Length Day 28, n=56, 58 | -1.434 (6.7887) | 0.485 (6.6552)
  FRC Diameter Day 12, n=56, 59 | -0.247 (1.8777) | 0.059 (1.1657)
  FRC Diameter Day 28, n=56, 58 | -0.261 (1.8672) | -0.047 (1.1522)
  TLC Length Day 12, n=58, 59 | 0.295 (4.0608) | -0.663 (3.8027)
  TLC Length Day 28, n=56, 59 | 0.168 (4.5501) | -0.495 (3.7295)
  TLC Diameter Day 12, n=58, 59 | -0.067 (1.0127) | -0.056 (0.5098)
  TLC Diameter Day 28, n=56, 59 | -0.046 (1.0240) | -0.082 (0.5579)
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 2.89, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.04, 95% CI 2-sided [1.00 to 1.07] — FRC Length Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 8.49, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.99 to 1.05] — FRC Length Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 86.21, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.02, 95% CI 2-sided [0.98 to 1.07] — FRC Diameter Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 75.20, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.98 to 1.05] — FRC Diameter Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 5: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 84.29, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.97 to 1.01] — TLC Length Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 6: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 71.08, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.98 to 1.01] — TLC Length Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 7: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 34.93, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.98 to 1.01] — TLC Diameter Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 8: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 25.05, Bayesian repeated measures model — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.98 to 1.01] — TLC Diameter Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval

7. Secondary Outcome: Change From Baseline in Imaging Trachea Length/Diameter After 12 Days of Treatment and After 28 Days of Treatment
Description: Imaging trachea length/diameter was derived from HRCT to evaluate the effect of once daily inhaled dose of GSK2269557 on lung parameters. TLC is the volume in the lungs at maximal inflation and FRC is the volume in the lungs at the end-expiratory position. The Baseline for the assessment on Day 12 and Day 28 is the Screening value. Change from Baseline is the post-Baseline value minus the Baseline value. The change from Baseline data is presented for Day 12 and Day 28 for trachea length/diameter. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 12 and Day 28
Population: ITT Population excluding the subject with a pacemaker.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- GSK2269557 1000 µg: Participants received 1000 µg of GSK2269557 two inhalations per day administered via a dry powder inhaler for a duration of 84 days.
Arm/Group | Placebo | GSK2269557 1000 µg
Number analyzed (Participants) | 62 | 63
ratio
  FRC Length/Diameter Day 12, n=56 | -0.030 (0.7717) | 0.000 (0.5620)
  FRC Length/Diameter Day 28, n=56 | -0.017 (0.7469) | 0.059 (0.5169)
  TLC Length/Diameter Day 12, n=5 | 0.024 (0.3602) | -0.023 (0.2913)
  TLC Length/Diameter Day 28, n=5 | 0.004 (0.3715) | -0.006 (0.2783)
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Superiority or Other; p = 28.51, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.97 to 1.06] — FRC Length/Diameter Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Superiority or Other; p = 32.15, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.01, 95% CI 2-sided [0.97 to 1.05] — FRC Length/Diameter Day 28. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 3: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Superiority or Other; p = 66.51, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 0.99, 95% CI 2-sided [0.97 to 1.02] — TLC Length/Diameter Day 12. The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval
Statistical Analysis 4: Comparison: Placebo vs GSK2269557 1000 µg; Test type: Superiority or Other; p = 45.28, Bayesian repeated measures model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Posterior Median Ratio = 1.00, 95% CI 2-sided [0.98 to 1.03] — TLC Length/Diameter Day 28 The data entered to the 95% confidence interval represents the 95% equi-tailed credible interval

8. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events were collected from the start of study treatment until the follow-up contact.
Time Frame: From start of IP through the Study Phase (84 days post-dose) (assessed up to follow-up duration of approximately 100 days)
Population: All Subjects Population: all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Participants | 41 | 49

9. Secondary Outcome: Number of Participants With Abnormal Hematology Parameters
Description: Hematology parameter included Hematocrit (HCT), Hemoglobin (HB), Lymphocytes (LC), Platelet Count (PC), Total Neutrophils (TN), and White Blood Cell (WBC) count at the indicated timepoints: Day 1, Day 12, Day 28, Day 56, Day 84, and at follow-up/Early withdrawal. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Day 1, Day 12, Day 28, Day 56, Day 84 and at follow-up (approximately 100 Days)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Participants
  High HCT Screening/Day 1, n=63, 62 | 4 | 1
  High HCT Day 12, n=60, 58 | 1 | 1
  High HCT Day 28, n=57, 58 | 1 | 1
  High HCT Day 56, n=55, 52 | 1 | 0
  High HCT Day 84, n=49, 53 | 2 | 1
  High HCT Follow-up/Early Withdraw, n=54, 53 | 4 | 0
  High HB Screening/ Day 1, n=63, 63 | 0 | 1
  High HB Day 12, n=60, 58 | 0 | 0
  High HB Day 28, n=57, 58 | 0 | 0
  High HB Day 56, n=55, 52 | 0 | 0
  High HB Day 84, n=49, 53 | 0 | 0
  High HB Follow-up/Early Withdraw, n=54, 53 | 0 | 0
  Low LC Screening/ Day 1, n=62, 60 | 9 | 7
  Low LC Day 12, n=59, 58 | 2 | 2
  Low LC Day 28, n=56, 57 | 3 | 3
  Low LC Day 56, n=54, 52 | 2 | 0
  Low LC Day 84, n=48, 50 | 2 | 0
  Low LC Follow-up/Early Withdraw, n=53, 53 | 1 | 1
  High PC Screening/Day 1, n=63, 63 | 0 | 0
  High PC Day 12, n=58, 57 | 0 | 0
  High PC Day 28, n=57, 58 | 1 | 0
  High PC Day 56, n=55, 52 | 0 | 0
  High PC Day 84, n=49, 53 | 0 | 0
  High PC Follow-up/Early Withdraw, n=54, 53 | 0 | 0
  Low PC Screening/ Day 1, n=63, 63 | 0 | 0
  Low PC Day 12, n=58, 57 | 0 | 0
  Low PC Day 28, n=57, 58 | 0 | 0
  Low PC Day 56, n=55, 52 | 0 | 0
  Low PC Day 84, n=49, 53 | 0 | 0
  Low PC Follow-up/Early Withdraw, n=54, 53 | 0 | 0
  Low TN Screening/ Day 1, n=62, 60 | 0 | 0
  Low TN Day 12, n=59, 58 | 0 | 1
  Low TN Day 28, n=56, 57 | 0 | 0
  Low TN Day 56, n=54, 52 | 0 | 0
  Low TN Day 84, n=48, 50 | 0 | 0
  Low TN Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  High WBC Screening/ Day 1, n=63, 63 | 0 | 1
  High WBC Day 12, n=56, 56 | 0 | 1
  High WBC Day 28, n=56, 57 | 0 | 0
  High WBC Day 56, n=54, 52 | 0 | 0
  High WBC Day 84, n=48, 50 | 0 | 0
  High WBC Follow-up/Early Withdraw, n=53, 53 | 0 | 2
  Low WBC Screening/ Day 1, n=63, 63 | 0 | 0
  Low WBC Day 12, n=56, 56 | 0 | 0
  Low WBC Day 28, n=56, 57 | 0 | 0
  Low WBC Day 56, n=54, 52 | 0 | 0
  Low WBC Day 84, n=48, 50 | 0 | 0
  Low WBC Follow-up/Early Withdraw, n=53, 53 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters
Description: Clinical Chemistry parameters included Alanine Amino Transferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Calcium (Ca), Glucose, Potassium (K), Sodium (Na), and Total Bilirubin (TBL) at the indicated timepoints: Day 1, Day 12, Day 28, Day 56, Day 84, and at follow-up/Early withdrawal. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Day 1, Day 12, Day 28, Day 56, Day 84 and at follow-up (approximately 100 days)
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Participants
  High ALT Screening/ Day 1, n=63, 63 | 0 | 1
  High ALT Day 12, n=61, 60 | 0 | 0
  High ALT Day 28, n=58, 60 | 1 | 0
  High ALT Day 56, n=55, 56 | 0 | 0
  High ALT Day 84, n=52, 55 | 0 | 0
  High ALT Follow-up/Early Withdraw, n=53, 54 | 0 | 0
  Low Albumin Screening/ Day 1, n=63, 63 | 0 | 0
  Low Albumin Day 12, n=61, 60 | 0 | 0
  Low Albumin Day 28, n=58, 60 | 0 | 0
  Low Albumin Day 56, n=55, 56 | 0 | 0
  Low Albumin Day 84, n=52, 55 | 0 | 0
  Low Albumin Follow-up/Early Withdraw, n=53, 53 | 1 | 1
  High ALP Screening/ Day 1, n=63, 63 | 0 | 0
  High ALP Day 12, n=61, 60 | 1 | 0
  High ALP Day 28, n=58, 60 | 1 | 0
  High ALP Day 56, n=55, 56 | 0 | 0
  High ALP Day 84, n=52, 55 | 0 | 0
  High ALP Follow-up/Early Withdraw, n=53, 54 | 1 | 0
  High AST Screening/ Day 1, n=63, 63 | 0 | 1
  High AST Day 12, n=61, 60 | 0 | 0
  High AST Day 28, n=58, 60 | 0 | 0
  High AST Day 56, n=55, 56 | 0 | 0
  High AST Day 84, n=52, 55 | 0 | 0
  High AST Follow-up/Early Withdraw, n=53, 54 | 1 | 1
  High Ca Screening/ Day 1, n=63, 63 | 0 | 0
  High Ca Day 12, n=61, 60 | 0 | 0
  High Ca Day 28, n=58, 60 | 0 | 0
  High Ca Day 56, n=55, 56 | 0 | 0
  High Ca Day 84, n=52, 55 | 0 | 0
  High Ca Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  Low Ca Screening/ Day 1, n=63, 63 | 0 | 0
  Low Ca Day 12, n=61, 60 | 0 | 0
  Low Ca Day 28, n=58, 60 | 0 | 0
  Low Ca Day 56, n=55, 56 | 0 | 0
  Low Ca Day 84, n=52, 55 | 0 | 0
  Low Ca Follow-up/Early Withdraw, n=53, 53 | 0 | 1
  High Glucose Screening/ Day 1, n=63, 63 | 6 | 8
  High Glucose Day 12, n=61, 60 | 2 | 6
  High Glucose Day 28, n=58, 60 | 1 | 3
  High Glucose Day 56, n=55, 56 | 3 | 5
  High Glucose Day 84, n=52, 55 | 5 | 3
  High Glucose Follow-up/Early Withdraw, n=53, 53 | 4 | 6
  Low Glucose Screening/ Day 1, n=63, 63 | 0 | 0
  Low Glucose Day 12, n=61, 60 | 0 | 0
  Low Glucose Day 28, n=58, 60 | 0 | 0
  Low Glucose Day 56, n=55, 56 | 0 | 0
  Low Glucose Day 84, n=52, 55 | 0 | 0
  Low Glucose Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  High Potassium Screening/ Day 1, n=63, 63 | 1 | 1
  High Potassium Day 12, n=61, 60 | 2 | 0
  High Potassium Day 28, n=58, 60 | 2 | 0
  High Potassium Day 56, n=55, 56 | 0 | 0
  High Potassium Day 84, n=52, 550 | 0 | 0
  High Potassium Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  Low Potassium Screening/ Day 1, n=63, 63 | 0 | 0
  Low Potassium Day 12, n=61, 60 | 0 | 0
  Low Potassium V4 Day 28, n=58, 60 | 0 | 0
  Low Potassium Day 56, n=55, 56 | 0 | 0
  Low Potassium Day 84, n=52, 55 | 0 | 0
  Low Potassium Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  High Sodium Screening/ Day 1, n=63, 63 | 0 | 0
  High Sodium Day 12, n=61, 60 | 0 | 0
  High Sodium Day 28, n=58, 60 | 0 | 0
  High Sodium Day 56, n=55, 56 | 0 | 0
  High Sodium Day 84, n=52, 55 | 0 | 0
  High Sodium Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  Low Sodium Screening/ Day 1, n=63, 63 | 1 | 0
  Low Sodium Day 12, n=61, 60 | 1 | 0
  Low Sodium Day 28, n=58, 60 | 0 | 0
  Low Sodium Day 56, n=55, 56 | 0 | 0
  Low Sodium Day 84, n=52, 55 | 1 | 0
  Low Sodium Follow-up/Early Withdraw, n=53, 53 | 0 | 0
  High TBL Screening/ Day 1, n=63, 63 | 1 | 0
  High TBL Day 12, n=61, 60 | 0 | 0
  High TBL Day 28, n=58,60 | 0 | 0
  High TBL Day 56, n=55, 56 | 0 | 0
  High TBL Day 84, n=51, 55 | 0 | 0
  High TBL Follow-up/Early Withdraw, n=53, 54 | 1 | 1

11. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Vital signs included high and low diastolic and systolic blood presure (BP), and high and low heart rate (HR). Vital signs outside the range of potential clinical importance are presented at the indicated timepoints: Day 1, Day 12, Day 28, Day 56, Day 84, follow-up/Early withdrawal and at any visit post-baseline . Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Day 1, Day 12, Day 28, Day 56, Day 84 and at follow-up (approximately 100 days)
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Participants
  High DBP Screening/Day 1, n=63, 63 | 1 | 0
  High DBP Day 12, n=61, 60 | 0 | 0
  High DBP Day 28, n=58, 60 | 0 | 0
  High DBP Day 56, n=55, 56 | 1 | 0
  High DBP Day 84, n=52, 55 | 0 | 0
  High DBP Follow-up/Early Withdraw, n=55, 60 | 0 | 0
  High DBP Any Visit Post Baseline, n=62, 62 | 1 | 0
  Low DBP Screening/ Day 1, n=63, 63 | 0 | 0
  Low DBP Day 12, n=61, 60 | 1 | 0
  Low DBP Day 28, n=58, 60 | 0 | 0
  Low DBP Day 56, n=55, 56 | 0 | 0
  Low DBP V6 Day 84, n=52, 55 | 0 | 0
  Low DBP Follow-up/Early Withdraw, n=55, 60 | 0 | 0
  Low DBP Any Visit Post Baseline, n=62, 62 | 1 | 0
  High SBP Screening/ Day 1, n=63, 63 | 2 | 3
  High SBP Day 12, n=61, 60 | 0 | 1
  High SBP Day 28, n=58, 60 | 0 | 0
  High SBP Day 56, n=55, 56 | 2 | 1
  High SBP Day 84, n=52, 55 | 1 | 1
  High SBP Follow-up/Early Withdraw, n=55, 60 | 1 | 1
  High SBP Any Visit Post Baseline, n=62, 62 | 3 | 2
  Low SBP Screening/ V1 Day 1, n=63, 63 | 0 | 0
  Low SBP Day 12, n=61, 60 | 0 | 0
  Low SBP Day 28, n=58, 60 | 0 | 0
  Low SBP Day 56, n=55, 56 | 0 | 0
  Low SBP Day 84, n=52, 55 | 0 | 0
  Low SBP Follow-up/Early Withdraw, n=55, 60 | 0 | 0
  Low SBP Any Visit Post Baseline, n=62, 62 | 0 | 0
  High HR Screening/ Day 1, n=63, 63 | 0 | 2
  High HR Day 12, n=61, 60 | 0 | 0
  High HR Day 28, n=58, 60 | 2 | 2
  High HR Day 56, n=55, 56 | 0 | 1
  High HR Day 84, n=52, 55 | 0 | 1
  High HR Follow-up/Early Withdraw, n=55, 60 | 1 | 1
  High HR Any Visit Post Baseline, n=62, 62 | 2 | 3
  Low HR Screening/ Day 1, n=63, 63 | 0 | 0
  Low HR Day 12, n=61, 60 | 0 | 0
  Low HR Day 28, n=58, 60 | 0 | 0
  Low HR Day 56, n=55, 56 | 0 | 0
  Low HR Day 84, n=52, 55 | 0 | 0
  Low HR Follow-up/Early Withdraw, n=55, 60 | 0 | 0
  Low HR Any Visit Post Baseline, n=62, 62 | 0 | 0

12. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG)
Description: 12-lead ECG was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected using the Fridericia's formula (QTcF). Clinically non-significant (CN) and Clinically significant (CS) abnormal ECG measurements are presented for Day 1, Day 12, Day 28, Day 56, Day 84, follow-up/Early withdrawal and at any visit post-baseline. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Day 1, Day 12, Day 28, Day 56, Day 84 and at follow-up (approximately 100 days)
Population: All Subject Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Participants
  CN ECG Screening/ Day 1, n=63, 63 | 45 | 40
  CS ECG Screening/ Day 1, n=63, 63 | 0 | 0
  CN ECG Day 12, n=61, 60 | 43 | 40
  CS ECG Day 12, n=61, 60 | 0 | 0
  CN ECG Day 28, n=58, 60 | 41 | 40
  CS ECG Day 28, n=58, 60 | 1 | 1
  CN ECG Day 56, n=55, 56 | 36 | 39
  CS ECG Day 56, n=55, 56 | 1 | 0
  CN ECG Day 84, n=52, 55 | 36 | 38
  CS ECG Day 84, n=52, 55 | 1 | 0
  CN ECG Follow-up/Early Withdraw, n=56, 60 | 35 | 43
  CS ECG Follow-up/Early Withdraw, n=56, 60 | 1 | 0
  CN ECG Any Visit Post Baseline, n=63, 62 | 51 | 51
  CS ECG Any Visit Post Baseline, n=63, 62 | 3 | 1

13. Secondary Outcome: Day 1 Plasma Concentration up to 24 Hours (Hrs) Post-dose
Description: Plasma samples were collected at pre-dose, 5 minutes (min), 3 hrs, and 24 hrs post-dose on Day 1. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Pharmacokinetic (PK) Population: all participants in the Safety Population for whom a PK sample was obtained and analyzed. Safety Population comprises of all participants who were randomized.
Time Frame: Pre-dose, 5 min, 3 hrs and 24 hrs
Population: Pharmacokinetic (PK) Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GSK2269557 1000 mcg
Number analyzed (Participants) | 62
pg/mL
  Pre-dose, n=61 | 33.0 (NA) — Only 5 of the 61 values had not been imputed as zero; therefore, calculation of the SD would result in a potentially misleading value and hence is omitted from the data display (if >30% of values are imputed then the SD will not be included).
  5 min, n=60 | 476.6 (520.85)
  3 hrs, n=61 | 553.7 (326.98)
  24 hrs, n=20 | 539.0 (482.76)

14. Secondary Outcome: Trough Concentration After 12 Days, 28 Days, 56 Days and 84 Days of Treatment
Description: Trough concentrations are presented for Pre-dose Day 12, Pre-dose Day 28, Pre-dose Day 56, and Pre-dose Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Pre-dose Day 12, Day 28, Day 56, and Day 84
Population: PK Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GSK2269557 1000 mcg
Number analyzed (Participants) | 62
pg/mL
  Pre-dose Day 12, n=57 | 1001.8 (669.05)
  Pre-dose Day 28, n=60 | 1028.8 (798.38)
  Pre-dose Day 56, n=55 | 1119.8 (1389.53)
  Pre-dose Day 84, n=54 | 948.6 (1078.31)

15. Secondary Outcome: Changes From Baseline in Forced Expiratory Volume in One Second (FEV1) Measured Daily
Description: FEV1 is the volume of air that can forcibly be blown out in one second. A triplicate FEV1 measurement were taken daily in the morning before dose administration. Baseline is defined as the assessment on Day 1 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84.Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 28, and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
mL
  Day 28, n=55, 58 | -70.4 (43.07) | -72.2 (41.28)
  Day 84, n=46, 54 | -83.3 (49.73) | -22.7 (46.77)
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.487, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -2.0, 95% CI 2-sided [-118.5 to 115.3] — Day 28
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.816, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 60.6, 95% CI 2-sided [-73.3 to 194.3] — Day 84

16. Secondary Outcome: Changes From Baseline in Peak Expiratory Flow (PEF) Measured Daily
Description: PEF is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration. Baseline is defined as the assessment on Day 1 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84.Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 28, and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
L/min
  Day 28, n=54, 57 | -13.12 (60.421) | -4.76 (57.578)
  Day 84, n=45, 53 | -0.52 (65.374) | -0.85 (71.170)

17. Secondary Outcome: Percent Change From Baseline in Diffusion Capacity (DLco, Kco) After 28 Days and After 84 Days of Treatment
Description: DLco is diffusing capacity o f the lungs for carbon monoxide and is defined as the extent to which oxygen passes from the air sacs of the lungs into the blood. KCO is the carbon monoxide transfer coefficient. It is an index of the efficiency of alveolar transfer of carbon monoxide. Baseline is defined as the assessment on Day 2 and percent change from Baseline is the post-Baseline value minus Baseline value/100. Change from Baseline data is presented for Day 28 and Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Percent
  DLco Day 28, n=53, 56 | -2.783 (9.3950) | -0.687 (8.2655)
  DLco Day 84, n=45, 51 | -2.385 (9.6016) | 0.560 (9.5434)
  Kco Day 28, n=53, 55 | -2.745 (9.7851) | -0.875 (8.0041)
  Kco Day 84, n=45, 50 | -2.367 (10.2835) | -0.759 (8.7801)

18. Secondary Outcome: Change From Baseline in Total Lung Capacity (TLC) After 28 Days and After 84 Days of Treatment
Description: TLC is the maximum amount of air that can fill the lungs. Baseline is defined as the assessment on Day 2 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Note: values mentioned as 95% confidence interval below are in fact values of 95% credible interval.
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: L
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
L
  Day 28, n=53, 59 | -0.010 [-0.211 to 0.190] | -0.155 [-0.344 to 0.035]
  Day 84, n=47, 55 | -0.149 [-0.462 to 0.163] | -0.029 [-0.320 to 0.265]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.151, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.144, 95% CI 2-sided [-0.420 to 0.133] — Day 28
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.712, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.121, 95% CI 2-sided [-0.305 to 0.551] — Day 84

19. Secondary Outcome: Change From Baseline in Residual Volume After 28 Days and After 84 Days of Treatment
Description: Residual volume is a lung volume representing the amount of air left in the lungs after a forced exhalation. Baseline is defined as the assessment on Day 2 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Note: values mentioned as 95% confidence interval below are in fact values of 95% credible interval.
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: L
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
L
  Day 28, n=53, 59 | -0.157 [-0.441 to 0.129] | 0.022 [-0.249 to 0.292]
  Day 84, =47, 54 | -0.113 [-0.430 to 0.206] | 0.001 [-0.299 to 0.296]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.817, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.180, 95% CI 2-sided [-0.216 to 0.570] — Day 28
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.697, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.114, 95% CI 2-sided [-0.324 to 0.549] — Day 84

20. Secondary Outcome: Change From Baseline in Functional Residual Capacity After 28 Days and After 84 Days of Treatment
Description: Functional residual capacity is the volume of air present in the lungs at the end of passive expiration. Baseline is defined as the assessment on Day 2 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
L
  Day 28, n=52, 59 | 0.0010 (0.86637) | -0.0919 (0.92501)
  Day 84, =46, 55 | -0.2219 (1.06874) | -0.0505 (1.41910)

21. Secondary Outcome: Change From Baseline in Specific Resistance (sRaw) After 28 Days and After 84 Days of Treatment
Description: sRaw is the measure of specific resistance. Baseline is defined as the assessment on Day 2 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: KPa*s
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
KPa*s
  Day 28, n= 17, 17 | 0.9734 (0.45833) | 0.8372 (0.49176)
  Day 84, n=11, 13 | 0.9949 (0.24484) | 0.8495 (0.39565)

22. Secondary Outcome: Change From Baseline in Specific Conductance (sGaw) After 28 Days and After 84 Days of Treatment
Description: Baseline is defined as the assessment on Day 2 and change from Baseline is the post-Baseline value minus Baseline value. Change from Baseline data is presented for Day 28 and Day 84. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).Note: values mentioned as 95% confidence interval below are in fact values of 95% Credible Interval.
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: 1/KPA*S
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
1/KPA*S
  Day 28, n=47, 52 | 0.875 [0.773 to 0.990] | 1.024 [0.910 to 1.150]
  Day 84, =40, 47 | 0.965 [0.860 to 1.083] | 1.075 [0.967 to 1.197]
Statistical Analysis 1: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.965, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 1.171, 95% CI 2-sided [0.988 to 1.388]
Statistical Analysis 2: Comparison: Placebo vs GSK2269557 1000 mcg; Test type: Superiority or Other; p = 0.913, Bayesian repeated measures model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 1.114, 95% CI 2-sided [0.953 to 1.305]

23. Secondary Outcome: Questionnaires CAT and MMRC Scale at Baseline, Day 28 and Day 84
Description: The chronic obstructive pulmonary disease (COPD) assessement test (CAT) and Modified Medical Research Council (MMRC) Dyspnea Scale were completed at the indicated timepoints: Baseline, Day 28 and Day 84. CAT and MMRC scales are prestned as: 1.I never cough/I cough all the time 2.I have no phelgm in my chest at all/My chest is completely full of phelgm 3. My chest does not feel tight at all/My chest feels very tight 4.Walk up hilll or stairs not breathless/Walk up hill or stairs very breathless 5. Not limited doing any home activities/Very limited doing any home activities 6. Confident leaving home/No confident leaving home 7. I sleep soundly/I don't sleep soundly because of my lung condition and 8. I have lots of energy/I have no energy at all. Baseline is defined as the assessment on Day 1. Score 0 indicates not troubled with breathlessness to 4:too breathless. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Day 28 and Day 84
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Scores on a scale
  never cough/cough all the time D28, n=58, 60 | -0.4 (1.16) | -0.7 (1.14)
  never cough/cough all the time D84, n=53, 55 | -0.6 (1.48) | -0.7 (0.99)
  No phlegm/full of phlegm in chest D28, n=58, 60 | -0.6 (1.26) | -0.3 (1.24)
  No phlegm/full of phlegm in chest D84, n=53, 55 | -0.8 (1.20) | -0.6 (1.18)
  No tightness/very tight chest D28, n=58, 60 | -0.2 (1.30) | -0.3 (1.16)
  No tightness/very tight chest D84, n=53, 55 | -0.1 (1.43) | -0.3 (1.34)
  Hill/stairs nobreathless/breathlessD28, n=58, 60 | -0.5 (0.98) | -0.5 (1.08)
  Hill/stairs nobreathless/breathless D84, n=53, 55 | -0.4 (1.43) | -0.3 (1.03)
  Unlimited/limited home activity D28, n=58, 60 | -0.3 (1.43) | -0.3 (1.15)
  Unlimited/limited home activity D84, n=53, 55 | -0.3 (1.24) | -0.1 (1.39)
  Confident/not confident leave home D28, n=58, 60 | -0.4 (1.24) | -0.1 (1.27)
  Confident/not confident leave homeD84, n=53, 55 | -0.2 (1.49) | -0.3 (1.34)
  Sound sleep/No sound sleep D28, n=58, 60 | -0.4 (1.11) | -0.2 (1.30)
  Sound sleep/No sound sleep D84, n=53, 55 | -0.3 (1.60) | -0.3 (1.36)
  Lot of energy/no energy D28, n=58, 60 | -0.1 (1.46) | -0.3 (1.22)
  Lot of energy/no energy D84, n=53, 55 | -0.2 (1.49) | -0.3 (1.25)
  CAT Total Score D28, n=58, 60 | -2.9 (6.05) | -2.6 (5.13)
  CAT Total Score D84, n=53, 55 | -3.0 (7.16) | -3.1 (5.45)
  MMRC Dyspnoea Score D28, n=58, 60 | -0.4 (0.75) | -0.2 (0.72)
  MMRC Dyspnoea Score D84, n=53, 55 | -0.4 (0.95) | -0.3 (0.71)

24. Secondary Outcome: Number of Participants With Treatment Failures
Description: Treatment failure types are presented as: recurrent exacerbations, prolonged treatment of current exacerbation (beyond 14 days), additional treatment with systemic / oral corticosteroids and / or antibiotics, and requirement for invasive mechanical ventilation.
Time Frame: 13 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2269557 1000 mcg
Number analyzed (Participants) | 63 | 63
Participants
  Recurrent exacerbation | 17 | 13
  Prolonged Treatment of current exacerbation | 9 | 7
  continuation of treatment with SOC/antibiotics | 4 | 3
  Additional treatment with SOC/antibiotics | 6 | 6
  Requirement of invasive mechanical ventilation | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication up to approximately 100 days.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of investigational product.
Arm/Group | Placebo | GSK2269557 1000 mcg
Serious Adverse Events (participants affected / at risk) | 10/63 | 8/63
Other Adverse Events (participants affected / at risk) | 15/63 | 31/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | GSK2269557 1000 mcg (N=63)
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | GSK2269557 1000 mcg (N=63)
Dry mouth (Gastrointestinal disorders) | 5 | 2
Headache (Nervous system disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 22
Hypertension (Vascular disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.